# Project Title

Does rosuvastatin delay progression of atherosclerosis in people with HIV infection at moderate cardiovascular risk?

A multicentre, randomized, double blind, placebo-controlled trial

Version Date: 14/02/2014 Version Number: 2.2

## **INVESTIGATORS**

Professor Jennifer Hoy (PI)

Dr Janine Trevillyan

Professor Suzanne Crowe

Dr Julian Elliott

A. Professor Anthony Jaworowski

Dr James Shaw

**Professor Anthony Dart** 

The Alfred Hospital

Monash University

Melbourne Australia

#### Contact:

Infectious Diseases Department

Alfred Hospital

55 Commercial Road

Melbourne VIC 3004

PO Box 315 Prahran

Victoria 3181 Australia

Telephone: 03 90762000

Fax: 03 90766557

## INVESTIGATORS SWITZERLAND

Dr Alexandra Calmy (PI and person responsible according to art. 7 Oclin for the study conduct in Switzerland)

Prof François Mach (Cardiology)

Dr Baris Gencer (Cardiology)

Dr Roman Sztajzel (Neurology)

Employees:

Rachel Spycher Elbes (Coordinator)

Cecile Delhumeau (Statistician)

## Contact of PI:

Infectious Diseases Department / HIV Unit (coordinating centre for Swiss sites)
Hôpitaux Universitaires de Genève
4, rue Gabrielle Perret Gentil
CH-1211 Genève 14
Switzerland

Telephone: +41 (0)22 372 98 12

Fax: +41 (0)22 372 98 20

| "] | l'a | bl | e | of | Con | ten | ts |
|----|-----|----|---|----|-----|-----|----|

| 1 | Si | gnature Form | 6 |
|----|------|-------------------------------------------------|----|
| 2 | Li | st of abbreviations | 7 |
| 3 | D | efinition of Terms | 8 |
| 4 | Pr | rotocol Synopsis | 9 |
| 5 | Fl | ow Chart | 11 |
| 6 | Ва | ackground | 12 |
| | 6.1 | Relationship between HIV infection and CVD | 12 |
| | 6.2 | Surrogate markers of cardiovascular outcomes | 13 |
| | 6.3 | Statin therapy | 13 |
| | 6.4 | Selection of doses | 14 |
| | 6.5 | Rationale for performing study | 14 |
| | 6.6 | Sample size | 14 |
| | 6.7 | Hypothesis | 15 |
| 7 | St | udy objectives | 15 |
| | 7.1 | Primary Objective | 15 |
| | 7.2 | Secondary Objectives | 15 |
| 8 | St | udy Design | 16 |
| | 8.1 | Design | 16 |
| | 8.2 | Duration | 17 |
| | 8.3 | Study centres | 17 |
| 9 | St | udy Population | 17 |
| | 9.1 | Inclusion Criteria | 17 |
| | 9.2 | Exclusion criteria. | 17 |
| | 9.3 | Prohibitions | 18 |
| | 9.4 | Removal of participants from therapy/assessment | 18 |
| | 9.5 | Pregnancy | 19 |
| 1( | 0 | Study Medication | 19 |
| | 10.1 | Rosuvastatin | 19 |
| | 10.2 | Placebo | 19 |
| | 10.3 | Packaging and Labelling | 19 |
| | 10.4 | Timing of dosing | 20 |
| | 10.5 | Storage | 20 |
| | 10.6 | Drug Accountability | 20 |
| | 10.7 | Compliance assessment | 20 |
| | 10.8 | Warnings and precautions | 20 |

| 10.9 | Concomitant medications | 21 |
|-------|----------------------------------------------|----|
| 10. | 9.1 Contraindications | 21 |
| 10. | 9.2 Warfarin | 21 |
| 10. | 9.3 Antiretrovirals | 21 |
| 10.10 | Drug interactions list | 22 |
| 10.11 | Blinding and Emergency Unblinding | 23 |
| 11 A | Assessments | 23 |
| 11.1 | Calculations | 24 |
| 11.2 | Laboratory Assessments | 25 |
| 11.3 | Carotid IMT | 26 |
| 11.4 | Pulse Wave Velocity | 27 |
| 12 V | isit Schedule | 27 |
| 12.1 | Screening | 27 |
| 12. | 1.1 Eligibility | 28 |
| 12.2 | Inclusion Criteria | 28 |
| 12.3 | Exclusion criteria | 28 |
| 12.4 | Randomisation | 29 |
| 12.5 | Baseline visit | 29 |
| 12.6 | Week 12 visit | 30 |
| 12.7 | Week 24 visit | 30 |
| 12.8 | Week 48 visit | 30 |
| 12.9 | Week 72 visit | 31 |
| 12.10 | Week 96 visit | 31 |
| 12.11 | Unscheduled visits | 32 |
| 12.1 | Withdrawal visit | 32 |
| 12.2 | Time windows | 32 |
| 13 A | Adverse Events | 32 |
| 14 S | erious Adverse Events | 33 |
| 14.1 | Serious Adverse Event Reporting Requirements | 33 |
| 15 E | Oata safety and monitoring board | 34 |
| 16 T | rial or site discontinuation | 35 |
| 17 S | tatistical Analysis | 35 |
| 18 I | nsurance and Finances | 36 |
| 19 ( | Quality Control and quality assurance | 36 |
| 19.1 | Source documents | 36 |
| 19.2 | Retention of essential documents | 36 |

| 19.3 | Data protection | 37 |
|-------|-----------------------------------------------------------|----|
| 19.4 | Monitoring, audits and inspections | 37 |
| 20 Pu | ablications and presentations | 37 |
| 21 R | eferences | 38 |
| 22 A | ppendix | 41 |
| 22.1 | Case Record Forms | 41 |
| 22.1 | .1 Screening Visit | 41 |
| 22.1 | .2 Baseline Visit | 47 |
| 22.1 | .3 Week 12 Visit | 48 |
| 22.1 | .4 Week 24 Visit | 49 |
| 22.1 | .5 Week 48 Visit | 50 |
| 22.1 | .6 Week 72 Visit | 52 |
| 22.1 | .7 Week 96 Visit | 53 |
| 22.1 | .8 Unscheduled Visits | 55 |
| 22.2 | Serious Adverse Event (SAE) Form | 56 |
| 22.3 | Units of measurement and reference ranges | 57 |
| 22.4 | Units of measurement and reference ranges for Swiss sites | 59 |
| 22.5 | Patient Informed Consent Form | 61 |
| 22.6 | Severity Grading of Adverse Events | 74 |

# 1 Signature Form

**Phone** 

I, the undersigned, have reviewed this Protocol, including Appendices. I will conduct the clinical study as described and I will adhere to GCP/ICH and all the local ethical and regulatory requirements.

| Principal Investigator Melbourne (AUS) | Signature | Date |
|---|---|---|
| Title | | |
| Institution and address | | |
| Phone | | |
| <b>Principal Investigator Geneva (CH)</b><br>Dre Alexandra Calmy | Signature | Date |
| <b>Title</b><br>MD, PD médecin adjoint agrégé | | |
| <b>Institution and address</b><br>Consultation des maladies infectieuses / uni<br>Hôpitaux Universitaires de Genève. 4, rue C | | 1 Genève 14 |
| <b>Phone</b><br>+41 22 372 98 12 | | |
| For additional Swiss sites: | | |
| Site Name: | | |
| Site main investigator | Signature | Date |
| Title | | |
| Institution and address | | |

#### 2 List of abbreviations

ACCF American College of Cardiology Federation

AE Adverse Events

AHA American Heart Association

AIDS Acquired immunodeficiency syndrome

Alb Albumin

ALP Alkaline phosphatase
ALT Alanine aminotransferase
AMI Acute Myocardial Infarction
ART Antiretroviral Therapy

ARV Antiretroviral BMI Body Mass Index

Ca Calcium

cART Combination Antiretroviral Therapy

CD4+ cells CD4+ T-cell count CHD Coronary Heart Disease

cIMT Carotid artery Intima Media Thickness

Cl Chloride

CMV Cytomegalovirus

CPK Creatinine phosphokinase

cPWV Carotid-femoral pulse wave velocity

Cr Creatinine

CrCl Creatinine Clearance
CRF Case Report Form
CVA Cerebrovascular accident
CVD Cardiovascular disease
CVE Cardiovascular events
D.A.D -RS D.A.D risk score

D.A.D. Data collection on Adverse events of anti-HIV Drugs

DBP Diastolic Blood Pressure

DSMB Data Safety and Monitoring Board

ECG Electrocardiograph

eGFR estimated glomerular filtration rate ESC European Society of Cardiology

FBE Full Blood Examination FRS Framingham Risk Score

GGT Gamma- glutamyl transpeptidase HaCH HIV and Cardiovascular Health

Hb Haemoglobin HCO<sub>3</sub> Bicarbonate

HDL-C High-density lipoprotein cholesterol HIV Human Immunodeficiency Virus

HMG Co-A 3-hydroxy-3-methylglutaryl coenzyme A

HUG Geneva University Hospitals hsCRP High sensitivity C-reactive protein

K+ Potassium

LDL-C Low-density lipoprotein cholesterol

LFT Liver Function Tests

LPS Lipopolysaccharide Lymp Lymphocyte Count

MAC Mycobacterium avian complex

MDRD Modification of Diet in Renal Disease

Na Sodium

Neut Neutrophil Count

PBMC Peripheral blood mononuclear cells
PBS Pharmaceutical Benefits Scheme
PCP Pneumocystis jirovecii pneumonia

Plt Platelets

PML Progressive multifocal leucoencephalopathy

PO<sub>4</sub> Phosphate

PVD Peripheral vascular disease

RNA Ribonucleic acid

SAE Serious Adverse Events
SBP Systolic Blood Pressure
SHCS Swiss HIV Cohort Study

SLE Systemic Lupus Erythematosus Statin HMG Co-A reductase inhibitor

TC Total Cholesterol
TG Triglycerides

TIA Transient ischaemic attack

TP Total Protein

UEC Urea, Electrolytes and Creatinine

ULN Upper limit of normal

Ur Urea

VAS Visual Analogue Scale

VIDRL Victorian Infectious Diseases Reference Laboratory

WCC Total White Cell Count WHF World Health Federation

β-HCG Beta-human chorionic gonadotropin

## 3 Definition of Terms

Study medication the medication under investigation (rosuvastatin) or the corresponding

placebo product administered for blinding

## 4 Protocol Synopsis

**Protocol title:** Does rosuvastatin delay progression of atherosclerosis in people with HIV infection at moderate cardiovascular risk? A randomized, placebo-controlled trial

**Primary Objective:** The primary objective is to determine the effect of rosuvastatin on atherosclerosis progression in individuals with HIV infection who are at moderate cardiovascular risk.

**Study Design:** This study will be a randomized, double blinded, placebo controlled, multicentre trial comparing the effect of rosuvastatin 20mg daily versus placebo over 96 weeks in people with HIV infection who are at moderate cardiovascular risk (as estimated by a Framingham Risk Score (FRS) between 10 - 15%). Participants will be randomised 1:1 to active rosuvastatin 20mg once daily or matching placebo. Participants on a protease inhibitor will receive dose reduced rosuvastatin (10 mg).

**Planned sample size:** 102 HIV positive participants (72 participants in Melbourne and 30 in Switzerland)

#### **Inclusion Criteria**

- 1. Provision of written, informed consent
- 2. Age >30 years
- 3. Moderate coronary heart Disease (CHD) risk, defined as FRS of 10-15%1
- 4. HIV positive
- 5. Stable ARV regimen > 3 months (i.e. no recent drug change [changes in dosages are accepted])
- 6. Plasma HIV viral load <200copies/ml for  $\ge 6$  months

#### **Exclusion criteria**

- 1. Recommended use of lipid lowering drug therapy according to Australian Guidelines (National heart foundation 2012)2
- 2. Family History of myocardial infarction or stroke
- 3. Type 2 Diabetes
- 4. Familial hypercholesterolemia
- 5. Aboriginal or Torres Strait Islander people with LDL-C >2.5 mmol/L
- 6. Blood pressure  $\geq 180/110$
- 7. Documented history of:
  - a. Ischemic stroke or transient ischemic attack (TIA)
  - b. Peripheral arterial disease
  - c. Congestive heart failure
  - d. Coronary artery disease or ECG findings consistent with prior MI
- 8. Carotid artery stenosis or >50% occlusion of the carotid artery
- 9. Total Cholesterol > 7.5 mmol/L
- 10. Triglyceride level >4.0 mmol/L
- 11. HDL-c <1 and Total cholesterol > 6.5 mmol/L
- 12. Current or prior (last 6 months) statin, ezetimibe, fibrate or niacin therapy

- 13. Contraindication to statin use
  - a. Pregnancy or lactation
  - b. Hypersensitivity to statins
  - c. Known myopathy or baseline CK > 3x ULN
  - d. Contraindicated concurrent medication
  - e. Current cyclosporine, fusidic acid or oral corticosteroid use
- 14. Concomitant antiplatelet drug
- 15. Unable to complete study procedures
- 16. Any active, clinically significant disease
- 17. Concomitant renal or hepatic disease, defined as the presence of the following:
  - a. Creatinine Clearance <50ml/min
  - b. Transaminase (ALT, AST) above 3 times upper normal limit
  - c. Acute hepatic failure
  - d. Compensated cirrhosis Child Class B or C

## **Study procedures**

Carotid intima media thickness (cIMT), carotid-femoral pulse wave velocity (cPWV) and biomarkers of immune activation and inflammation will be measured at baseline and compared to values obtained after 48 and 96 weeks of treatment with the study medication. Other procedures will include assessments of safety, fasting lipid and glucose analysis and storage of plasma and peripheral blood mononuclear cells (PBMCs) for future research.

## 5 Flow Chart

| Assessment | Screen | Baseline | e Post randomization | | | | |
|---|---|---|---|---|---|---|---|
| Week | -4 | 0 | 12 | 24 | 48 | 72 | 96 |
| Written Informed consent | X | | | | | | |
| Inclusion / exclusion criteria | X | | | | | | |
| Demographic questionnairea | X | | | | | | |
| Physical examination b | X | X | | | X | | X |
| Compliance assessmente | | | | | X | | X |
| Weight & Height measurementa | X | | | | X | | X |
| Adverse event assessmente | | X | X | X | X | X | X |
| Risk Score Calculations | X | | | | | | |
| <b>Laboratory Assessments</b> | | | | | | | |
| T Cells | X | | X | X | X | X | X |
| HIV RNA viral load | X | | X | X | X | X | X |
| FBEg | X | X | X | X | X | X | X |
| Biochemistryh | X | X | X | X | X | X | X |
| Fasting Lipids/glucosei | X | X | | X | X | | X |
| hsCRP | | X | X | | | | X |
| Research Blood samples j | | X | X | | X | | X |
| Structural assessments | | | | | | | |
| Carotid IMT <sub>k</sub> | X | | | | X | | X |
| Pulse Wave Velocity | X | | | | X | | X |

- <sup>a</sup> Demographic data, medical history and medication questionnaire (will be performed with a trained interpreter if required)
- b Includes blood pressure measurement, cardiovascular examination; electrocardiogram (ECG) at screening visit only
- $_{\mbox{\scriptsize c}}$  See appendix17.2: Compliance self-assessment questionnaire and visual analogue scale
- d Height will only be measured at screening visit. Body Mass Index (BMI) will be calculated at screening and 12 and 24 month post randomisation
- e Unscheduled visits may be performed for safety/tolerability concerns
- f Framingham (FRS) and Data Collection on Adverse Events of Anti-HIV Drugs (D.A.D) risk scores calculated g Full Blood Examination: Haemoglobin, White cell count, Lymphocyte count, Neutrophil count, Platelet count h Including sodium, potassium, bicarbonate, chloride, calcium, phosphate, urea, creatinine; Liver function tests (LFTs): alanine aminotransferase (ALT), alkaline phosphatase (ALP), total protein, albumin; creatinine phosphokinase (CPK), pregnancy screen in women with child bearing potential
- i Participants will fast overnight and have bloods taken in the morning for total cholesterol (TC), low-density lipoprotein cholesterol (LDL), high-density lipoprotein cholesterol (HDL), triglycerides (TG) and glucose j Blood for markers of innate immunity and inflammation; see Section11.2 for full description of testing to be performed and stored bloods for future projects
- k Carotid intima media thickness (cIMT) will be performed on the left and right common carotid arteries, 12 consecutive measurements will be made 1-3cm proximal to the carotid bulb in areas identified as being without plague.
- <sup>1</sup> Carotid-femoral Pulse Wave Velocity (cPWV) will be determined by using simultaneous applanation tonometry of the carotid and femoral arteries. Only for Australian site.

## 6 Background

## 6.1 Relationship between HIV infection and CVD

#### HIV positive patients have a two-fold increased risk of CVD

cART has dramatically reduced HIV-related morbidity and mortality resulting in a rapidly growing population of older patients living with HIV<sub>3,4</sub>. The major burden of illness, health care utilization and premature death in people with HIV is now due to diseases of ageing, particularly CVD, which occurs not only at higher rates (2 fold increased relative risk)s but also at a younger age than in the general population<sub>6</sub>. In a case-control study performed at the Alfred Hospital (AH) in 2010, the incidence of cardiovascular events (CVE) in HIV positive people was 8.5 cases per 1000 person years<sub>7</sub>, twice the rate reported rates in HIV negative males of similar age (3.9 per 1000 person years)<sub>8</sub>. HIV may promote atherogenesis by a reduction in high-density lipoprotein cholesterol (HDL-C) and reverse cholesterol transport<sub>9</sub>, immune activation and inflammation, increases in thrombosis and fibrinolysis and endothelial dysfunction<sub>10,11</sub>.

Cardiovascular risk is likely to be underestimated in people with HIV. The contributing effect of HIV-associated immune activation and cART on CVD risk in HIV positive people is not considered in traditional CVD risk scores (such as the FRS<sub>1</sub>). In a cohort study conducted by our group at the AH, the FRS correlated only moderately with carotid intima media thickness (cIMT), a well validated surrogate marker of CVE. 11% of HIV positive patients with low (<10%) FRS had a cIMT >0.7 mm (*HIV and cardiovascular health (HaCH) study pilot data)*. Whilst others have also shown the true CVD risk is likely to be underestimated by FRS in people with HIV<sub>12</sub>, correlation between FRS and risk of CVD in HIV patients remains uncertain.

#### CVD is associated with immune activation and inflammation in people with HIV.

The increased risk of CVD in HIV positive people is thought to be due to a combination of the effects of HIV infection, toxicity from ART and conventional CVD risk factors. The Data collection on Adverse Effects of Anti-HIV Drugs (D:A:D) study, (including data from the AH HIV cohort) provided the first evidence of increased incidence of myocardial infarction with longer duration of cART (26% increased rate of AMI per year of ART use)13, in addition to different relative risks according to class of ART used and specific ART drugs14,15. HIV infection is associated with chronic immune activation and inflammation that persists despite virologic suppression16. The increased risk of CVD decreases with successful ART, but does not return to that of the general population17. It is also known that increased levels of T cell activation in HIV positive participants predicts subclinical carotid artery disease18.

The pathogenesis of atherosclerosis is complex but inflammation is a key driving force. Inflammation drives oxidation of plasma low-density lipoprotein (LDL-C) and activates endothelial cells allowing monocytes to attach to them via their CD11b receptor and then migrate into the forming atherosclerotic plaque within the vessel wall. Bacterial endotoxin or lipopolysaccharide (LPS) is a potent inducer of inflammation; chronic endotoxemia and high plasma soluble CD14 (sCD14, released from monocytes and macrophages) are found in most HIV positive people. This is secondary to HIV-induced CD4+ T-cell depletion in the gut and loss of mucosal integrity allowing translocation of microbial products (e.g. LPS) across the gut19. LPS binds to monocytes via CD14, signalling cellular activation and pro-inflammatory

cytokine (e.g. IL-6) production that is critical for the initiation of CVD. Production of CRP in the liver is primarily driven by IL-6, which activates further IL-6 production by monocytes<sub>20</sub>.

## 6.2 Surrogate markers of cardiovascular outcomes

Given the large number of patients that have been required to perform clinical outcome studies in CVD it is neither feasible nor practical to design such a study in the HIV population. Thus surrogate markers of CVD endpoints are necessary to allow to effects of therapeutic interventions on CVD risk to be assessed in this population. In this study we will be utilising two well validated surrogate markers of CVD; cIMT and cPWV.

#### Carotid intima media thickness

cIMT has been validated as an independent predictor of CVD outcomes in the general population after adjustment for other risk factors21. cIMT has been used as an endpoint in clinical trials evaluating the effect of statins on CVD outcomes with a correlation between treatment induced reductions in cIMT and AMI22. Several cross-sectional studies have shown HIV+ people have greater cIMT than age and sex matched controls23-25, and significantly higher progression rates than historical reports in HIV negative populations.

## **Pulse Wave Velocity**

cPWV is a surrogate measure of arterial stiffness and is considered a marker of atherosclerosis. It has been shown to be an independent predictor of CVD events in prospective studies26. Increased arterial stiffness has been reported in HIV infection compared with HIV negative controls25,27,28. Rosuvastatin has been shown to improve aortic arterial stiffness with changes strongly correlated with reduction in LDL29. cPWV will not be performed at Swiss sites.

## **6.3** Statin therapy

Statins are HMG-CoA reductase inhibitors that lower total cholesterol, improve endothelial function, and halt progression of atherosclerosis<sup>30</sup>. Randomized trials of rosuvastatin in the general population have shown a reduction in major CVD events and in the inflammatory biomarker high sensitivity C-reactive protein (hsCRP) in healthy adults with normal LDL levels (the JUPITER trial)<sup>31</sup>. High levels of baseline hsCRP were an independent predictor of CVD in this cohort<sup>32</sup>. The absolute CVD event reduction with rosuvastatin was greatest in those with highest baseline hsCRP levels and in those who achieve low hsCRP levels regardless of LDL level achieved<sup>33,34</sup>. The cIMT effect size seen with statin therapy correlates with reduction in LDL and baseline cIMT<sup>30</sup>. As previously shown HIV positive people have, on average, greater cIMT and faster cIMT progression rates, thus it is likely that the magnitude of effect seen with statin therapy may be greater.

Furthermore, statins are immune modulators, and inhibit inflammation in part by reducing chemokine and pro-inflammatory cytokine synthesis by monocytes, inhibiting monocyte adhesion to the blood vessel wall as well as improving the function of other cells involved in atherogenesis (smooth muscle cells, platelets, endothelial cells)35-37. Rosuvastatin is predicted to alter the plasma levels of inflammatory markers and monocyte phenotype by week 12. Atorvastatin decreased CRP, IL-6 and CCL2 levels in 4-6 weeks in HIV negative participants38,39. Rosuvastatin has been shown to induce a 16% reduction in hsCRP in stable ART-treated HIV positive participants over 45 days40. High dose atorvastatin over 8 weeks in ART naive HIV positive participants resulted in significant decreases in immune activation (CD4+ HLA-DR+, CD8+ HLA-DR+ and CD8+ CD38+ T cells)41. These effects may provide

additional benefit in HIV positive participants given high baseline levels of immune activation and inflammation and the association between these markers and CVD outcomes.

#### 6.4 Selection of doses

The Jupiter study, using a rosuvastatin dose of 20 mg daily, demonstrated reductions in LDL cholesterol by 50% and hsCRP by 37%; resulting in a 50% reduction in vascular events<sup>31</sup>. The METEOR study reported a significant reduction in cIMT progression after 12 months of rosuvastatin therapy with the divergence continuing to increase with further follow-up out to 24 months<sup>22</sup>. Most rosuvastatin (90%) is excreted unchanged, while 10% undergoes limited metabolism by cytochrome P450 2C9. Pharmacokinetic studies of drug-drug interactions in healthy volunteers have shown that protease inhibitors (PI) in current use caused a 2.4-4.7 fold increase in Cmax and 1.5-3 fold increase in AUC for rosuvastatin<sup>42,43</sup>. For the participants receiving a non-PI based cART regimen, a dose of 20 mg rosuvastatin (1 x20 mg tablet) will be used. Participants on any PI-based cART regimen will receive 1 X 10 mg rosuvastatin (effective exposure 20 mg daily).

## 6.5 Rationale for performing study

The key questions regarding CVD in HIV positive people is the extent to which the pathogenesis of CVD differs between HIV positive people and the general population, and whether treatment thresholds established in the general population for the initiation of conventional CVD interventions (such as statin therapy) apply to HIV positive people. Given the role of inflammation in atherosclerosis, strong evidence of higher cIMT and greater progression rates of cIMT in HIV infection it is plausible that HIV positive people may experience a clinical benefit from the earlier initiation of statin therapy.

This study will prospectively collect validated surrogate CVD endpoint data and extensive biomarker investigations in HIV positive participants, enabling controlled comparisons of these endpoints between the two treatment arms. It is likely that HIV positive patients at moderate FRS (who would not normally qualify for stain therapy on current guidelines) will experience quantifiable benefits from administration of rosuvastatin due either to higher baseline levels of atherosclerosis not reflected in FRS or due to differential immunological effects in the unique milieu of immune activation seen in HIV positive people.

## 6.6 Sample size

The METEOR study of rosuvastatin in HIV negative participants with low to intermediate CVD risk found a mean Common Carotid Artery cIMT progression rate of 0.0088 mm/2 years in the placebo arm and 0.0004mm/2 years in the rosuvastatin arm22, giving an effect size of 0.0084 mm/2 years (95% relative reduction) with a standard deviation (SD) of 0.033 mm/year. A pilot study in HIV positive patients at the AH (n=10) found that in participants treated with non-nucleoside reverse transcriptase inhibitors (the most common cART regimen), the mean cIMT progression rate was 0.04 mm/year with a SD of 0.0782 mm (personal communication Dmitri Sviridov, Baker IDI), similar to estimated values proposed for cIMT progression in HIV positive participants at low to intermediate CVD risk (mean 0.045 mm/year, SD 0.08 mm; 62).

Conservatively assuming a cIMT progression rate of 0.080 mm with a SD of 0.09 mm over 2 years and near stabilisation of cIMT (95% relative reduction) with rosuvastatin, we can assume an effect size of 0.076 mm with a SD of 0.09 mm. Sample size was calculated using an independent groups t-test with an alpha threshold of 1% and a power of 90%. Based on these hypotheses, with 44 participants in each group this study will be able to detect an effect

size of 0.076 mm with a SD of 0.09 mm over 2 years between the 2 groups. With an estimated 15% total drop-out rate over 96 weeks, we estimate that a total study population of 102 will be required.

## 6.7 Hypothesis

That treatment with rosuvastatin 20mg daily will delay progression of atherosclerosis and reduce biomarkers of activation and inflammation in HIV positive people with intermediate FRS.

## 7 Study objectives

## 7.1 Primary Objective

The primary objective is to determine the effect of rosuvastatin on atherosclerosis progression in individuals with HIV infection who are at moderate cardiovascular risk.

The primary outcome measure will be the difference in cIMT progression (measured as a change from baseline) between the rosuvastatin and placebo arms.

## 7.2 Secondary Objectives

Secondary objectives are to determine in HIV positive patients:

- 1. The safety profile of rosuvastatin
- 2. The effect of rosuvastatin on vessel wall function and biomarkers of atherosclerosis and innate immune activation
- 3. The effect of rosuvastatin on fasting lipids and glucose
- 4. Whether baseline measures of immune activation and inflammation predicts cIMT or progression of cIMT
- 5. Whether a change in measures of immune activation and inflammation from baseline after three months of rosuvastatin therapy predicts progression of cIMT

Secondary outcome measures include:

- 1. The rate of adverse effects (symptomatic and biochemical) between the two treatment arms
- 2. The effect of rosuvastatin on cIMT and cPWV
- 3. The effect of rosuvastatin on immunological and inflammatory markers (including sCD14, sCD163, neopterin, S-VCAM-1, adiponectin, CCL2, inflammatory (CD16+) monocyte expression of CD38, CX3CR1 and CD11b)
- 4. The effect of rosuvastatin on fasting total cholesterol, LDL, HDL, TG and glucose levels after 6, 12 and 24 months of therapy
- 5. The relationship between baseline measures of sCD14, sCD163, and neopterin and baseline cIMT
- 6. The relationship between baseline measures of sCD14, sCD163, and neopterin and rate of progression of cIMT
- 7. The relationship between change from baseline to 3 months in markers of immune activation and inflammation (sCD14, CCL2, and inflammatory (CD16+) monocyte phenotypic expression of CD38, CD11b) and progression of cIMT at 12 and 24 months.

## 8 Study Design

#### 8.1 Design

The study will be a randomized, double blinded, placebo controlled, multicentre trial comparing the effect of rosuvastatin 20 mg daily versus placebo over 96 weeks in people with HIV infection at moderate cardiovascular risk.



Individuals (n=102) with moderate CVD risk, as estimated by the FRS (10-15% 10 year risk of CVD), who do not qualify for statin therapy under Australian guidelines2, will be randomized 1:1 to active rosuvastatin 20mg once daily or matching placebo.

Placebo and rosuvastatin capsules identical in shape and colour will be used to help preserve blinding. Participants on a protease inhibitor based cART regimen will receive 10 mg rosuvastatin or matching placebo.

#### Randomisation

A computerized random number generator will be used to assign treatment arms. Block Randomisation will be stratified by country.

There will be seven study visits over the 96 week duration of the study.

cIMT, cPWV and biomarkers of immune activation and inflammation will be

measured at screening visit and compared to values obtained after 48 and 96 weeks of treatment with the study medication.

cIMT and cPWV measurements will be performed in duplicate, by the same operator at the AH Heart Centre or the Swiss site, who will remain blinded to participant randomization, throughout the study.

All samples will be processed on site at the AH or the Swiss site. Standard laboratory assessments (i.e. biochemistry, full blood examination (FBE), fasting lipids, hsCRP) will be processed by AH pathology department or the Swiss sites' local laboratories. Markers of innate immunity and inflammation will be performed in the Burnet laboratories. Plasma and PBMCs will be separated from research bloods samples, frozen to -140oC and stored onsite in the Burnet laboratory for possible further analysis in the future.

For Switzerland: Plasma samples for testing of inflammation markers will be stored on site at minus 80° and shipped to central biobank (sérothèque) HUG for analysis at the HUG cardiology laboratory.

#### 8.2 Duration

Ninety-six (96) weeks per patient Expected duration for entire project – 5 years

## 8.3 Study centres

Patients will be recruited and followed at the Alfred Hospital (Victorian HIV service) Infectious Diseases Clinic.

Switzerland: Patients will be recruited within the HIV Cohort Network, at the following hospitals following regulatory approval: University Hospitals in Geneva, Lausanne, Berne, Zurich and Basel and the Cantonal Hospitals of St Gallen and Lugano, providing that these centers and affiliated Ethics Committee do accept to enrol patients in the present study. The patients will be recruited during their routine visits to the sites by the local investigators. The use of recruitment advertisements or flyers is not intended.

## 9 Study Population

#### 9.1 Inclusion Criteria

- 1. Provision of written, informed consent
- 2. Age >30 years
- 3. Moderate coronary heart Disease (CHD) risk, defined as FRS of 10-15%1
- 4. HIV positive
- 5. Stable ARV regimen > 3 months (i.e. no recent drug change [changes in dosages are accepted])
- 6. Plasma HIV viral load <200copies/ml for  $\ge 6$  months

#### 9.2 Exclusion criteria

- 1. Recommended use of lipid lowering drug therapy according to Australian Guidelines (National heart foundation 2012)2
- 2. Family History of myocardial infarction or stroke in a male first degree relative before 55 years of age, or a female first degree relative before 65 years of age
- 3. Type 2 Diabetes
- 4. Familial hypercholesterolemia
- 5. Aboriginal or Torres Strait Islander people with LDL-C > 2.5 mmol/L
- 6. Blood pressure  $\geq 180/110$
- 7. Documented history of:
  - a. Ischemic stroke or transient ischemic attack (TIA)
  - b. Peripheral arterial disease (regardless of severity)
  - c. Congestive heart failure
  - d. Coronary artery disease or ECG findings consistent with prior MI
- 8. Carotid artery stenosis or >50% occlusion of the carotid artery known previously or discovered during screening procedures
- 9. Total Cholesterol > 7.5 mmol/L
- 10. Triglyceride level >4.0 mmol/L
- 11. HDL-c <1 and Total cholesterol > 6.5mmol/L
- 12. Current or prior (last 6 months) statin therapy

- 13. Current or prior (last 6 months) use of ezetimibe
- 14. Current or prior (last 6 months) use of fibrates or niacin
- 15. Contraindication to statin use
  - a. Pregnancy or lactation
  - b. Hypersensitivity to statins
  - c. Known myopathy or baseline CK > 3x ULN
  - d. Contraindicated concurrent medication
  - e. Current cyclosporine, fusidic acid or oral corticosteroid use
- 16. Concomitant antiplatelet drug (Aspirin, Abciximab, Anagrelide, Cilostazol, Clopidogrel, Dipyridamole, Eptifibatide, Ticagrelor, Ticlopidine, Tirofiban, Terutroban)
- 17. Unable to complete study procedures (i.e. attendance at AH for cIMT and cPWV testing or cIMT images not accepted for analysis despite redo examination)
- 18. Any active, clinically significant disease (including but not limited to; pancreatitis, significant psychiatric disorders, acquired immunodeficiency syndrome (AIDS) defining illnesses) which may impact on the results of the study, increase the risk of serious adverse events (SAE) or limit participants life expectancy to < 24 months
- 19. Concomitant renal or hepatic disease, defined as the presence of the following:
  - a. Creatinine clearance <50 ml/min (calculated using the Cockroft-Gault equation)45
  - b. Transaminase (ALT, AST) above 3 times upper normal limit
  - c. Acute hepatic failure
  - d. Compensated cirrhosis Child Class B or C

#### 9.3 Prohibitions

Concurrent participation in non-related clinical trials is allowed as long as there is no impact on the objectives of this trial.

## 9.4 Removal of participants from therapy/assessment

Participants will be withdrawn from the trial if:

- 1. A SAE occurs which is thought to be related to involvement in the study
- 2. The subject withdraws consent
- 3. The subject becomes pregnant
- 4. The subject is diagnosed with clinical cardiovascular disease
  - a. Cardiovascular
    - i. Acute myocardial infarction (AMI)
    - ii. Development of angina
    - iii. New ECG changes consistent with cardiovascular disease
  - b. Cerebrovascular
    - i. Stroke or Transient Ischaemic Attack (TIA)
  - c. Peripheral vascular disease
    - i. Symptomatic claudication
- 5. The subject is diagnosed with an acute serious medical illness that would be a contraindication to statin therapy i.e.
  - a. Acute viral hepatitis (A, B or C)
- 6. CK or transaminase elevation (> 3 times)

7. Subject is judged by the investigator to be at significant risk of failing to comply with the provisions of the protocol so as to cause harm to self or seriously interfere with the validity of the study result.

## 9.5 Pregnancy

Women of child-bearing potential will be screened for pregnancy on admission to the study. Due to a lack of study data relating to the effects of statins on pregnant woman and/or the foetus those who are found to be pregnant will be excluded from study participation and referred to an appropriate medical service<sup>46</sup>.

Female participants will be advised to avoid pregnancy while participating in the study. Women who become pregnant after randomisation will be withdrawn from the trial but will continue to be monitored for the development of adverse events (AE) or serious adverse events (SAE).

For Switzerland: Women of childbearing potential must use two reliable contraceptive methods during the entire trial, from day 1 to one month after the end of the trial. Accepted methods are hormonal methods such as the birth control pill associated with a barrier method such as the preservative.

## **10 Study Medication**

Participants will be randomly assigned in a 1:1 ratio to receive rosuvastatin or matched placebo.

#### 10.1 Rosuvastatin

Rosuvastatin is a hypolipidaemic agent and member of the drug class of statins used to treat high cholesterol and related conditions. Rosuvastatin is licensed by the Australian Therapeutic Goods Administration (TGA) for the prevention of major cardiovascular events and in patients with hypercholesterolemia (including familial hypercholesterolemia). Rosuvastatin should be used as an adjunct to dietary modification.

Rosuvastatin capsules of 10mg and 20mg dosages will be purchased from the manufacturer - Astra Zeneca.

#### 10.2 Placebo

A placebo identical in appearance to rosuvastatin will be produced by Pharmaceutical Packaging Professionals (PPP)in Thebarton South Australia. Stability tests will be performed by PPP and lot numbers and expiry dates provided to the sites.

## 10.3 Packaging and Labelling

Packaging and labelling will be in accordance with the applicable local regulatory requirements.

The study medication will be packed into bottles by Pharmaceutical Packaging Professionals (PPP) and shipped to the sites.

Labels will contain the following information: "for clinical trial use only"; study name and number; lot number, expiry date or re-testing date; patient ID or randomization number; "keep out of reach of children"; storage condition; name of PI and Institution.

The study medication will be distributed to the patient by the local research investigator or study nurse.

## 10.4 Timing of dosing

Rosuvastatin is taken once daily and can be taken with or without food. Participants will be encouraged to take it at the same time every day with a glass of water. Catch up doses should NOT be taken in the setting of a missed/forgotten dose.

## 10.5 Storage

The study medication should be stored in its provided packaging at room temperature (<30°C) away from heat and moisture.

## 10.6 Drug Accountability

The Investigator is responsible for ensuring accountability for the study medication, including reconciliation of drugs and maintenance of drug records.

Drug accountability documentation will be performed according to the local regulatory requirements and will include confirmation of the study medication received at the site; the study medication distributed to the patient and returned by the patient; lost or destroyed study medication; corresponding dates, quantities, batch numbers, expiry dates, as well as subject identification numbers.

The investigator should maintain records that adequately document:

- That the subjects were provided the doses specified by the protocol/amendment(s)
- That all study medication provided to the site was fully reconciled.

## 10.7 Compliance assessment

Compliance to the study medication (rosuvastatin and placebo) will be assessed by self-reported questionnaire using a modified Medication Adherence Self-Report Inventory and visual analogue scale (VAS) 47.

If it appears that a participant is not taking the study medication according to protocol they will be counselled by the investigator in an attempt to improve compliance.

## 10.8 Warnings and precautions

#### Musculoskeletal reported side effects

HMG-CoA reductase inhibitors (statins) have been associated with rare cases of severe myopathy and rhabdomyolysis, accompanied by increases in creatine kinase (>10x upper normal limit), myoglobinuria, proteinuria, and renal failure, mainly observed in 40mg daily dosage. Concomitant use with gemfibrozil (fibric acid derivatives), niacin, cyclosporine, erythromycin (macrolides) or azole antifungals may increase the incidence and severity of musculoskeletal side effects. Milder forms of myotoxicity (i.e., myalgia) are commonly reported and occur in approximately 5% to 7% of patients taking a statin drug.

## Other reported side effects

frequent ( $\geq 1/100$ , <1/10):

- Myalgia
- Diabetes (JUPITER study 2,8% in the rosuvastatin arm versus 2,3% in the placebo arm)
- Headache, dizziniess

- Abdominal pain, constipation, nausea
- Asthenia

Occasional ( $\geq 100/10$ , < 1/10):

- Pruritis, rash

Rare ( $\geq 1/10'000$ ,  $\leq 1/1000$ ) side effets include:

- Myopathy, arthralgia
- Hepatic transaminases elevations
- Hypersensitivity reactions
- Pancreatitis

Very rare (<1/10'000) side effects:

- Jaundice, hepatitis
- Hematuria
- Polyneuropathy

Frequency unknown:

- Cough, dyspnea
- Diarrhea
- Steven-Johnson syndrome
- Necrotic myopathy
- Gynecomastia
- Oedema

## **10.9 Concomitant medications**

Participants are not to commence any new medication without notifying the study coordinators to allow an assessment for potential interactions with the study medication.

#### 10.9.1 Contraindications

The use of rosuvastatin is contraindicated in combination with the following medications. A patient requiring commencement of these medications following enrolment will be withdrawn from the study.

- Cyclosporine
  - o Combined uses significantly increases rosuvastatin exposure.
- Gemfibrozil and other fibrates
  - Combined use increases the risk of adverse skeletal muscle effects and should only be used with caution
- Niacin
  - Combined use increases the risk of adverse skeletal muscle effects and should only be used with caution
- Fusidic acid
  - Combined use increased rosuvastatin levels and the risk of adverse skeletal muscle effects

#### 10.9.2 Warfarin

Combined use of coumarin anticoagulants with rosuvastatin is not contraindicated but will lead to prolonged INR. Patients should have a stable INR prior to starting rosuvastatin. INR monitoring should occur at increased frequency upon initiation or alteration of rosuvastatin dose.

#### 10.9.3 Antiretrovirals

Participants must be on a stable ARV regimen for > 3 months (with HIV viral load <200 for >6 months) to be eligible for acceptance into the study. ARV regimens will remain at the

discretion of the patients treating physician who will be blinded to study medication but not involvement in the study.

Participants on any PI-based cART regimen will receive 1 x 10 mg rosuvastatin (effective exposure 20 mg daily).

Participants who require a change in antiretroviral regimen following randomisation on the basis of treatment failure or intolerability (that could not be attributed to the study medication) may remain within the study.

- Patients who switch from a PI containing regimen to a non-PI containing regimen will have the dose of rosuvastatin (or placebo) increased to 20mg daily
- Patients who switch from a non-PI containing regimen to a PI containing regimen will have the dose of rosuvastatin (or placebo) reduced to 10mg daily
- Switches within classes of ARV require no change in study medication dose

## 10.10 Drug interactions list<sub>m</sub>

Table below: Influence of concomitantly administered drugs on exposure to rosuvastatin (AUC, Cmax in descending order of effect size) based on published clinical trials. Source: Swiss Compendium (www.compendium.ch)

| Interacting Drug, dosage and treatment period | Rosuvastatin-dosage and treatment period | Effect on rosuvastatin AUC | Effect on rosuvastatin-Cmax |
|---|---|---|---|
| Ciclosporin 75 mg b.i.d. up to 200 mg b.i.d., 6 Months | 10 mg q.d., 10 days | 7,1 fold ↑ | 11 fold ↑ |
| Atazanavir 300 mg/Ritonavir<br>100 mg q.d., 8 days | 10 mg, single dose | 3,1 fold ↑ | 7 fold ↑ |
| Lopinavir 400 mg/Ritonavir<br>100 mg B.I.D., 17 days | 20 mg q.d., 7 days | 2,1 fold ↑ | 5 fold ↑ |
| Gemfibrozil 600 mg b.i.d., 7 days | 80 mg, single dose | 1,9 fold ↑ | 2,2 fold ↑ |
| Eltromobopag 75 mg q.d. ,<br>10 days | 10 mg, single dose | 1,6 fold ↑ | 2 fold ↑ |
| Darunavir 600 mg/Ritonavir<br>100 mg b.i.d., 7 days | 10 mg q.d., 7 days | 1,5 fold ↑ | 2,4 fold ↑ |
| Tipranavir 500 mg/Ritonavir<br>200 mg b.i.d., 11 days | 10 mg, single dose | 1,4 fold ↑ | 2,2 fold ↑ |
| Dronedaron 400 mg b.i.d. | No data | 1,4 fold ↑ | No data |
| Itraconazol 200 mg q.d., 5 days | 10 mg or 80 mg,<br>single dose | 1,4 fold ↑ | 1,4 fold ↑ |
| Ezetimibe 10 mg q.d., 14 days | 10 mg q.d., 14 days | 1,2 fold ↑ | 1,2 fold ↑ |
| Fosamprenavir 700 mg/<br>Ritonavir<br>100 mg b.i.d., 8 days | 10 mg, single dose | ↑ 8% | 1,5 fold ↑ |
| Aleglitazar 0,3 mg, 7 days | 40 mg, 7 Days | $\leftrightarrow$ | 1,1 fold ↑ |
| Silymarin 140 mg t.i.d., 5 days | 10 mg, single dose | $\leftrightarrow$ | $\leftrightarrow$ |
| Fenofibrat 67 mg t.i.d., 7 days | 10 mg, 7 Days | ↑ 7% | 1,2 fold ↑ |
| Rifampicin 450 mg q.d., 7 days | 20 mg, single dose | $\leftrightarrow$ | $\leftrightarrow$ |

m Source: Swiss Compendium and translated into the English by the Swiss site: www.compendium.ch

| Interacting Drug, dosage and treatment period | Rosuvastatin-dosage and treatment period | | Effect on rosuvastatin-Cmax |
|---|---|---|---|
| Ketoconazol 200 mg b.i.d., 7 days | 80 mg, single dose | ↑ 2% | $\leftrightarrow$ |
| Fluconazol 200 mg q.d., 11 days | 80 mg, single dose | ↑ 14% | $\leftrightarrow$ |
| Erythromycin 500 mg q.i.d., 7 days | 80 mg, single dose | 28%↓ | 31% ↓ |
| Baicalin 50 mg t.i.d., 14 Days | 20 mg, Single dose | 47%↓ | 19%↓ |

<sup>«↑»:</sup> Increase.

«↔»: No change (defined as <20% change of rosuvastatin -AUC, C-max).

## 10.11 Blinding and Emergency Unblinding

The personnel involved in the conduct of the trial as well as the study participants will remain blinded to the assigned study medication, throughout the trial.

Unblinding: The study physician may decide to break the randomization code of the participant for security reasons only. Emergency code breaking instructions will be provided to the sites. In Switzerland: the coordinating centre must be informed immediately if a code has been broken.

#### 11 Assessments

All assessments including screening and unplanned study visits will be recorded on the case report form (CRF) – See Appendix 22.1

## Demographic data, medical history and medication questionnaire

Patients will be questioned on details necessary for determining eligibility for entry into the trial and important study variables. Topics to be covered include, age, gender, race, presence of CVD risk factors (smoking status, family history of CVD etc.), past medical history, current medications and the presence of any allergies.

The questionnaire will be completed by a study investigator at the screening visit. At all subsequent visits patients will be asked:

- 1. If they have developed or been diagnosed with any new medical illnesses since the last review
- 2. If they have started or stopped any non-study medications
- 3. Their current smoking status.

#### **Compliance assessment**

1. Compliance with the study medication will be performed at two time points (Weeks 48 and 96) to estimate compliance throughout the study. A self-assessment question sheet and VAS will be used asking participants to estimate compliance over the last fortnight and month. (See appendix 22.2)

#### Physical examination

Consists of:

- 1. Complete physical examination
- 2. Blood pressure measurement with patient sitting

<sup>«↓»:</sup> Decrease.

- 3. Recording presence of bilateral lower limb peripheral pulses of the posterior tibial and the dorsalis pedis arteries
- 4. Anthropometry
  - a. Weight will be measured in kilograms (kg) with patient clothed; footwear removed
  - b. Height will be measured in metres (m) with footwear removed
  - c. Waist circumference (adapted from the International Diabetes Federation guidelines on the diagnosis and management of the metabolic syndrome)48
    - i. Subject should be standing erect dressed in underwear; all outer clothing should be removed.
    - ii. Make sure the tape does not compress the tissues during the measurement.
    - iii. Record the measurement after the subject has exhaled with the tape measure in a horizontal plane, midway between the inferior margin of the ribs and the superior border of the iliac crest.

## Electrocardiogram (ECG)

ECG will be performed by trained study investigators at screening visit.

All ECGs will be read by a blinded study doctor; all important abnormalities on the ECG will be reported. Specifically the presence of findings consistent with prior myocardial infarction (as defined by the 2007 Joint European Society of Cardiology/American College of Cardiology Federation/American Heart Association/World Health Federation (ESC/ACCF/AHA/WHF) Task Force49;

- Any Q-wave in leads  $V_2$ - $V_3 \ge 0.02$ s or QS complex in leads  $V_2$  and  $V_3$
- Q-wave  $\geq 0.03$ s and  $\geq 0.1$ mV deep or QS complex in leads I, II, aVL, aVF or V4-V6, in any two leads of a contiguous lead grouping (I, aVL, V6; V4-V6; II, III, aVF)
- R-wave  $\geq$  0.04s in V<sub>1</sub>-V<sub>2</sub> and R/S  $\geq$  1 with a concordant positive T-wave in the absence of a conduction defect

#### Adverse event assessment

See sections 13 and 14 for details on AE and SAE reporting and assessment At each study visit patients will be asked to report any untoward medical occurrences and will also be specifically questioned regarding the presence of:

- Myopathic symptoms (weakness, muscle pain)
- Gastrointestinal disturbance (diarrhoea, nausea, vomiting, abdominal pain)
- Jaundice

#### 11.1 Calculations

## Framingham Risk Score

Ten-year risk of developing "hard" coronary heart disease endpoints (myocardial infarction and coronary death) will be calculated based on the Framingham Risk Score using an online calculator available at www.old.mdcalc.com/framingham-coronary-heart-disease-risk-score-si-units/

#### **D.A.D Risk Score**

The D.A.D equation is a cardiovascular risk assessment model that is tailored for use in HIV positive participants, taking into account exposure to specific PIs, family history of CHD and previous, as well as current smoking status 50. A D.A.D. risk score will be calculated on all

participants at baseline to allow for a comparison with the FRS and to compare each measure with cIMT. The calculation will be performed using an online tool available at: http://www.cphiv.dk/tools/dadriskequations/tabid/437/default.aspx

## **Body Mass Index (BMI)**

A BMI will be calculated at screening visit and at the forty-eight (48) and ninety-six (96) week visits. Height will only be measured at screening and assumed to remain stable through the study period

BMI = Weight (kg) / height2 (m)

#### Creatinine clearance

An estimated creatinine clearance will be calculated at screening visit to determine eligibility for entry into the trial using the Cockroft-Gault equation45

For men 
$$Cl = \frac{1.23 \times \text{weight (kg)} \times (140 - age(years))}{\text{Creatinine ($\mu$mol/L)}}$$
For women  $Cl = \frac{1.03 \times \text{weight (kg)} \times (140 - age(years))}{\text{Creatinine ($\mu$mol/L)}}$ 

# 11.2 Laboratory Assessments

## Handling of Biological samples

All biological samples (excluding those for storage and testing of innate immunity) will be processed at the Alfred Hospital laboratory or the Swiss site; local laboratory reference ranges will apply (see appendix 22.3 and 22.4).

Biological samples for testing of innate immunity will be handled at the Burnet Institute. Plasma will be separated and frozen (-80°C). Plasma markers will be analysed on batched frozen samples by ELISA.

Swiss sites will store plasma samples (6mls per visit) at -80°C and ship to the HUG cardiology laboratory for testing of plasma markers. Innate immunity markers (PBMC) will not be performed at Swiss sites.

A separate laboratory SOP will be provided to all the Swiss sites.

#### **HIV** specific testing

HIV monitoring (CD4+ T-cell count and HIV viral load) will be performed at screening, baseline and weeks 12, 48, 72 and 96

## Laboratory assessments for safety

Routine laboratory assessments for safety and tolerability will be performed including:

- Full Blood Examination (FBE)
  - Consisting of; Haemoglobin (Hb), total White Cell Count (WCC),
     Lymphocyte Count (Lymp), Neutrophil Count (Neut) and Platelet count (Plt)
- Biochemistry
  - Oconsisting of; Sodium (Na), Potassium (K+), Chloride (Cl), Bicarbonate (HCO<sub>3</sub>), Calcium (Ca), Phosphate (PO<sub>4</sub>), Urea (Ur), Creatinine (Cr) and creatinine phosphokinase (CPK)

- An estimated glomerular filtration rate (eGFR) based on the Modification of Diet in Renal Disease (MDRD)<sub>51</sub> equation is calculated electronically by the AH laboratory and will be recorded
- Liver Function Tests: Total Protein (TP), Albumin (Alb), Bilirubin (Bil),
   Alanine aminotransferase (ALT), Alkaline phosphatase (ALP) and Gamma-glutamyl transpeptidase (GGT)
- Pregnancy screen in women with child bearing potential (at screening visit);
   Beta Human chorionic gonadotrophin (β-HCG)

## **Fasting metabolic parameters**

Patients will be requested to attend the study visit having fasted overnight (for 12 hours). Definition of fasting: no food, caffeine or caloric drinks; free water is allowed and encouraged. Samples will be sent for TC, HDL, LDL, TG and glucose. Study participants and site investigators will be blinded to the results of metabolic testing

until the completion of the study. This is to prevent self-modification of lifestyle or diet in an attempt to normalise out-of-range results

#### Markers of Innate immunity and inflammation

Markers of Innate immunity and inflammation will be measured at baseline, and weeks 12, 48, and 96.

For participants recruited in Melbourne only: A panel of innate immune markers selected from HaCH including monocyte markers (CD14, CD16) of activation (CD38), of expression linked to migration, adhesion and progression of atherosclerotic plaque (CD11b, CX3CR1) will be performed.

In participants from both sites in plasma, markers of inflammation (IL6, sCD163) and monocyte activation / chemokine ligands (sCD14, neopterin, CCL2), S-VCAM-1 and adinopectin will be measured.

High sensitivity C-reactive protein (hsCRP) will be performed by the AH laboratory according to standard protocols

#### **Stored Samples**

4ml of plasma will be stored indefinitely for possible future testing and research for participants that give their consent. Storage samples will be collected at baseline and weeks 12, 48 and 96.

Samples will be stored at -80<sub>°</sub>C in the Burnet research laboratory and -80°C at the Swiss sites. Swiss sites will transfer the samples to the HUG central "sérothèque" for storage. Participants recruited from the Alfred Hospital will also have PBMC's stored at -140 in the Burnet research laboratory.

#### 11.3 Carotid IMT

The bilateral carotid artery will be assessed for cIMT by B Mode ultrasound using a Philips iE33 with 11 MHz linear transducer (Melbourne). The Swiss sites will be using the ultrasound machine tested and accepted by the core lab in Montréal following the Standard Operating Procedures for cIMT. The cIMT measurement is a painless and harmless non-invasive ultrasound procedure performed on patients' left and right common carotid arteries. The procedure takes 20 minutes to perform. The cIMT defined as the distance between lumen-intima interface and media-adventia interface is measured from the 2D high resolution digital images obtained using an automated border-detection algorithm. cIMT will be

determined on areas identified as without plaque by 12 consecutive measurements made 1-3 cm proximal to the carotid bulb, but the presence of plaques will be noted. All measurements will be performed in duplicate, by the same operator at the AH Heart Centre or the Swiss site, who will remain blinded to participant randomization, throughout the study.

Investigators and patients will not receive results from cIMT (or cPWV – see below) until the end of the study, unless a significant carotid plaque warranting further investigation and management is identified. Patients who are identified as having a significant plaque will be withdrawn from the study and referred to a cardiologist at the AH or the Swiss site for further assessment and management as necessary.

## 11.4 Pulse Wave Velocity

Australian site only: cPWV will be determined using simultaneous applanation tonometry of the carotid and femoral arteries. PWV will be calculated as manubrium sternum-to-femoral artery distance minus carotid artery-to-manubrium sternum distance divided by the time interval between the carotid and femoral pulses calculated from the upstroke of the systolic waveform (maximum of the second derivative). The cPWV will be reported as the average of pulse waves recorded over a 10 second period. It is a painless and harmless procedure that takes 20 min to perform by trained operators. The co-efficient of variation for this measurement is 5%.

#### 12 Visit Schedule

## 12.1 Screening

The screening procedures will be completed in one visit at the study site. Participants will present to the study site, having fasted from overnight for at least 12 hours (no food, caffeine or caloric drink; free water is encouraged).

Written informed consent will be obtained at screening visit by trained research staff (see Appendix 22.5 and 22.6). Participants will be informed in written and orally prior to the screening visit and given sufficient time for reflexion before signing the consent form.

#### Assessments

- 1. Demographic data, medical history and medication questionnaire to be completed
- 2. Full physical examination including:
  - a. Height and weight
  - b. Assessment of peripheral pulses
  - c. Blood pressure
  - d. ECG
- 3. Laboratory assessments
  - a. FBE and biochemistry
  - b. Beta HCG for all women of child bearing potential
  - c. Fasting metabolic assessment
  - d. HIV viral load and CD4+ T cell count (and percentage)
- 4. Structural assessments
  - a. cIMT
  - b. cPWV (\*Melbourne Participants only)
- 5. Calculations
  - a. BMI

- b. Creatinine clearance
- c. FRS
- d. D.A.D. risk score

#### 12.1.1 Eligibility

Clinical eligibility will be recorded based on the inclusion (1-6) and exclusion criteria (7-26) listed below.

#### 12.2 Inclusion Criteria

- 1. Provision of written, informed consent
- 2. Age >30 years
- 3. Moderate coronary heart Disease (CHD) risk, defined as FRS of 10-15%1
- 4. HIV positive
- 5. Stable ARV regimen > 3 months (i.e. no recent drug change [changes in dosages are accepted])
- 6. Plasma HIV viral load <200copies/ml for  $\ge 6$  months

#### 12.3 Exclusion criteria

- 7. Recommended use of lipid lowering drug therapy according to Australian Guidelines (National heart foundation 2012)2
- 8. Family History of myocardial infarction or stroke in a male first degree relative before 55 years of age, or a female first degree relative before 65 years of age
- 9. Type 2 Diabetes
- 10. Familial hypercholesterolemia
- 11. Aboriginal or Torres Strait Islander people with LDL-C > 2.5 mmol/L
- 12. Blood pressure  $\geq 180/110$
- 13. Documented history of:
  - a) Ischemic stroke or transient ischemic attack (TIA)
  - b) Peripheral arterial disease (regardless of severity)
  - c) Congestive heart failure
  - d) Coronary artery disease or ECG findings consistent with prior MI
- 14. Carotid artery stenosis or >50% occlusion of the carotid artery known previously or discovered during screening procedures
- 15. Total Cholesterol > 7.5 mmol/L
- 16. Triglyceride level >4.0 mmol/L
- 17. HDL-c <1 and Total cholesterol > 6.5mmol/L
- 18. Current or prior (last 6 months) statin therapy
- 19. Current or prior (last 6 months) use of ezetimibe
- 20. Current or prior (last 6 months) use of fibrates or niacin
- 21. Contraindication to statin use
  - f. Pregnancy or lactation
  - g. Hypersensitivity to statins
  - h. Known myopathy or baseline CK > 3x ULN
  - i. Contraindicated concurrent medication
  - j. Current cyclosporine, fusidic acid or oral corticosteroid use

- 22. Concomitant antiplatelet drug (Aspirin, Abciximab, Anagrelide, Cilostazol, Clopidogrel, Dipyridamole, Eptifibatide, Ticagrelor, Ticlopidine, Tirofiban, Terutroban)
- 23. Unable to complete study procedures (i.e. attendance at AH for cIMT and cPWV testing or cIMT images not accepted for analysis despite redo examination)
- 24. Any active, clinically significant disease (including but not limited to; pancreatitis, significant psychiatric disorders, acquired immunodeficiency syndrome (AIDS) defining illnesses) which may impact on the results of the study, increase the risk of serious adverse events (SAE) or limit participants life expectancy to < 24 months,
- 25. Any active, clinically significant disease (including but not limited to; pancreatitis, significant psychiatric disorders, acquired immunodeficiency syndrome (AIDS) defining illnesses) which may impact on the results of the study, increase the risk of serious adverse events (SAE) or limit participants life expectancy to < 24 months
- 26. Concomitant renal or hepatic disease, defined as the presence of the following:
  - a. Creatinine clearance <50 ml/min (calculated using the Cockroft-Gault equation)45
  - b. Transaminase (ALT, AST) above 3 times upper normal limit
  - c. Acute hepatic failure
  - d. Compensated cirrhosis Child Class B or C

If the patient fulfils all eligibility criteria (1-26 above) then a baseline visit will be booked. CRFs from participants assessed but found to be ineligible for inclusion in the study will be entered into the database recording the reason for ineligibility.

## 12.4 Randomisation

Patients will be block randomised in a 1:1 ratio to receive rosuvastatin or placebo. Randomisation will be stratified by centre.

#### 12.5 Baseline visit

Participants will be required to present to the study site having fasted overnight for at least 12 hours (no food, caffeine or caloric drinks; free water is encouraged)

Assessments performed:

- 1. Targeted physical examination and updated history, assessment for new concomitant medications
- 2. Adverse event assessment
- 3. Laboratory assessments
  - a. Biochemistry
  - b. Fasting metabolic assessment
  - c. hsCRP
  - d. Markers of innate immunity and inflammation
  - e. Storage of plasma and PBMCs (\*Melbourne participants only) for possible further analysis in the future

Patients will be provided with a three (3) month supply of the study medication and educated regarding possible clinical signs of potential adverse events (muscle ache, fever, abdominal pain, jaundice, rash); regardless of randomisation. Patients will also be provided with contact details for study co-ordinators in case of adverse event.

#### **12.6 Week 12 visit**

Participants will be required to present to the study site having fasted overnight for at least 12 hours (no food, caffeine or caloric drinks; free water is encouraged)

## Assessments performed:

- 1. Assessment for adverse events
- 2. Laboratory assessment for:
  - a. FBE
  - b. Biochemistry
  - c. hsCRP
  - d. Markers of innate immunity and inflammation
  - e. HIV Viral load and CD4+ T-cell count (and percentage)
- 3. Storage of plasma and PBMCs (\*Melbourne participants only) for possible future analysis

Patients provided with a further three (3) month supply of the study medication.

#### 12.7 Week 24 visit

Participants will be required to present having fasted overnight for at least 12 hours (no food, caffeine or caloric drinks; free water is encouraged)

Assessments performed:

- 1. Assessment for adverse events
- 2. Laboratory assessment for:
  - a. Biochemistry
  - b. Fasting metabolic assessment
  - c. HIV Viral load and CD4+ T-cell count (and percentage)

Patients will be provided with a six (6) month supply of the study medication

#### 12.8 Week 48 visit

Participants will be required to present having fasted overnight for at least 12 hours (no food, caffeine or caloric drinks; free water is encouraged).

Assessments performed:

- 1. Targeted physical examination and updated history, assessment for new concomitant medications
- 2. Weight recorded
- 3. Compliance assessment
  - a. Self-assessment questionnaire and VAS
- 4. Adverse event assessment
- 5. Laboratory assessments
  - a. Biochemistry
  - b. Fasting metabolic assessment
  - c. HIV Viral load and CD4+ T-cell count (and percentage)
  - d. Markers of innate immunity and inflammation
  - e. Storage of plasma and PBMCs (\*Melbourne participants only) for possible further analysis in the future
- 6. Calculations

- a. Creatinine clearance
- b. BMI
- 7. Structural assessments
  - a. cIMT
  - b. cPWV (\*Melbourne participants only)

Patients will be provided with a six (6) month supply of the study medication

#### 12.9 Week 72 visit

Fasting NOT required for this visit

Assessments performed:

- 1. Assessment for adverse events
- 2. Laboratory assessment for:
  - a. Biochemistry
  - b. HIV Viral load and CD4+ T-cell count (and percentage)

Patients will be provided with a six (6) month supply of the study medication

#### 12.10 Week 96 visit

Participants will be required to present to the AH having fasted overnight for at least 12 hours (no food, caffeine or caloric drinks; free water is encouraged).

Assessments performed:

- 1. Targeted physical examination and updated history, assessment for new concomitant medications
- 2. Weight recorded
- 3. Compliance assessment
  - a. Self-assessment questionnaire and VAS
- 4. Adverse event assessment
- 5. Laboratory assessments
  - a. FBE
  - b. Biochemistry
  - c. Fasting metabolic assessment
  - d. hsCRP
  - e. HIV Viral load and CD4+ T-cell count (and percentage)
  - f. Markers of innate immunity and inflammation
  - g. Storage of plasma and PBMCs (\*Melbourne participants only) for possible further analysis in the future
- 6. Calculations
  - a. Creatinine clearance
  - b. BMI
- 7. Structural assessments
  - a. cIMT
  - b. cPWV (\*Melbourne participants only)

Patients will be advised to cease study medication. Statin will be prescribed according to phycisian's assessment.

#### 12.11 Unscheduled visits

Unscheduled visits may be initiated by study co-ordinators and doctors, participants or treating physicians. All assessments made during unscheduled visits will be recorded on the CRF.

This visit may involve, but is not limited to, the following assessments; targeted medical review and physical examination, additional laboratory examination for safety reasons. SAE or AE visits may occur as unscheduled visits.

#### 12.1 Withdrawal visit

For participants that fulfil any of the withdrawal criteria above a withdrawal visit is performed if the participant agrees. All assessments made during the withdrawal visit can be recorded on the CRF (unscheduled visit). This visit will include, but is not limited to, a targeted medical review and physical examination, laboratory examination for safety reasons (chemistry and haematology), pregnancy test for women and study drug return. Tests performed can vary according to the judgement of the study physician.

Clinical or biological abnormalities perceived at the withdrawal visit will be followed at an interval decided by the study physician, until they are resolved or baseline values obtained.

Participants that withdraw from the study may be contacted by telephone at study end for vital status, unless they refuse and this is documented.

In Australia: In the event of withdrawal of consent by the participant, the Form for withdrawal of participants is completed.

#### 12.2 Time windows

The baseline visit will occur within four (4) weeks of screening to allow for laboratory assessments to be completed and FRS to be calculated confirming eligibility Study visits at weeks 12 and 24 have a visit window of  $\pm$ 14 days (to allow for scheduling of structural assessments and subject convenience). Study visits at weeks 48, 72 and 96 have a visit window of  $\pm$ 4 weeks.

#### 13 Adverse Events

An AE is defined as follows:

Any untoward medical occurrence in a clinical investigation subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Pre-existing or recurrent conditions that occur during the study should not be considered as AEs unless they change in frequency or severity.

All AEs that occur from the time the subject consents to participate in the study and throughout the duration of the study shall be recorded as an AE in the individuals CRF. At the final study visit (week 96) any ongoing adverse events deemed related to study drug will be followed up for a minimum of 30 days and until resolution.

In case a treatment interruption is needed during the treatment period in the event of a suspected toxicity, the subject will not automatically be withdrawn from the trial, as long as treatment interruption does not exceed 4 weeks.

AEs and SAEs will be categorised and recorded as per the modified Division of AIDS table for grading the Severity of Adverse Events (see Appendix 22.6). Causal relationship of AEs and SAEs to the trial and the study medication will also be assessed.

#### 14 Serious Adverse Events

A serious adverse event (SAE) is defined as follows:

Any adverse drug experience occurring at any dose that results in any of the following outcomes:

- Death
- Life-threatening situation (subject is at immediate risk of death)
- In-patient hospitalisation or prolongation of existing hospitalisation
- Persistent or significant disability/incapacity
- Congenital anomaly/birth defect in the offspring of a subject who received the study drug
- Other medically significant events that may not be immediately life-threatening or result in death or hospitalization, but based upon appropriate medical and scientific judgement, may jeopardize the subject or may require medical or surgical intervention to prevent one of the outcomes listed above.

## 14.1 Serious Adverse Event Reporting Requirements

The Principal Investigator and/or the project coordinator (coordinating center for Swiss sites) must be notified immediately (within 24 hrs of awareness of the event) regarding the occurrence of any SAEs.

The Principal Investigator and/or the study monitor (coordinating center for Switzerland) will report any SAE that fulfils the criteria for expedited reporting (unexpected and drug related events) to the appropriate regulatory authorities within the required reporting time frame. SAEs must also be reported to the approving ethics committee(s) as required by the ethics committee reporting procedures.

SAEs must be reported during a subject's participation in the study (whether receiving study medication or not) or within 30 days of receiving the last dose of study agent, whichever is longer.

Any SAE that is ongoing at the final study visit (week 96) will be followed until resolution or stabilisation (for those events that will not resolve).

For Switzerland: Safety reporting will be performed according to regulatory requirements detailed in the Overview of safety reporting procedures that is published on the Swissethics (Swiss association of Ethics Committees for clinical trials) website:

<a href="http://www.swissethics.ch/doc/templates/Overview\_safety\_AGEK\_dec11\_final.pdf">http://www.swissethics.ch/doc/templates/Overview\_safety\_AGEK\_dec11\_final.pdf</a>.

The coordinating centre Geneva must be reported to immediately by the study site in case of an SAE or SUSAR. The coordinating centre Geneva will report all drug related events (Adverse Drug Reactions) to Swissmedic in an annual update safety report. All SUSARS/SUSADRs (Suspected, unexpected Serious Adverse Drug Reaction) will be reported.

to Swissmedic within 7 days for fatal and/or life threatening ADRs, 15 days for all other reportable ADRs.

## 15 Data safety and monitoring board

An independent Data safety and monitoring board (DSMB) will be set up to monitor the safety of and efficacy in the participants enrolled in the trial. The DSMB will be chaired by A. Carr. Members will include one cardiologist from Switzerland (Proposition: R Lerch), one methodologist (Proposition: Prof Perneger), and one statistician from Australia (Proposition: T Spelman).

Data will be sent to the DSMB every 24 weeks. A summary of SAEs, grade 3/4 AEs and laboratory toxicities, and AEs leading to discontinuation will be provided on a monthly basis.

There will be a single, un-blinded, interim safety and efficacy analysis and review meeting after the last participants has completed 48 weeks of follow-up. The following data will be reviewed:

#### Safety data:

- Participant recruitment, accrual, retention, and withdrawal information
- Adverse events (AEs) and serious adverse events (SAEs)
- Clinical test results and laboratory values
- Vital signs and physical exam outcomes
- Participant questionnaires
- Study drug dose information
- Any other safety-supporting data requested by the DSMB

## Efficacy data

• cIMT data (primary endpoint measure)

Primary outcome measures (cIMT) and the first secondary outcome measure (adverse effects) will be analysed. Based on these analyses, the DSMB will make recommendations regarding the continuation, modification or termination of the trial.

#### Stopping rules:

The DSMB may recommend stopping of the trial for the following reasons:

- The data show a significantly increased risk of serious adverse effects in one of the treatment groups.
- On the basis of a positive efficacy result only when the data are truly compelling and the risk of a false positive conclusion is acceptably low. The trial will only be stopped for positive efficacy if a strong statistically and clinically significant difference in cIMT is seen between treatment arms.
- If interim data suggest that the product under study is of no benefit (no trend indicating superiority of the product), or that accrual rates are too low and/or that noncompliance is too great to provide adequate power for identifying the specified benefit, the DSMB may consider whether continuation of the study is futile and may recommend termination on this basis.

• It becomes clear that successful completion of the study is not feasible (e.g. there is an excess of patient dropout, missing data, lack of recruitment etc).

The DSMB may recommend modifications to individual stopping rules if additional safety concerns arise during from their continuing reviews of the study data.

#### 16 Trial or site discontinuation

The trial leaders (Principal Investigator in Melbourne and Geneva) reserve the right to discontinue the trial at any time for the following reasons:

- Emergence of safety of other information that could significantly affect the continuation of the trial;
- Failure to meet expected enrolment goals overall or at a particular trial site;
- Violation of GCP or the agreement of the investigator to conduct the trial appropriately.

## 17 Statistical Analysis

Baseline characteristics will be summarized using median (interquartile range) for quantitative variables and frequency and percentage for qualitative variables.

#### 1. Analysis of the primary endpoint:

To study rosuvastatin effect from baseline to week 96 on mean and / or of left and right maximal IMT progression, multi-levels, repeated measures, linear mixed-effects models adjusted for demographics and/or traditional CVD risk factors and centre (Melbourne, Geneva, Lausanne, Berne, Zurich, Basel, St. Gallen, Lugano) will be used. Levels used for the data will be patient and carotid artery locations (CCA, ICA, BIF and ECA) within patients; the repeated measure will be time (baseline, week 48 and week 96).

A comparison across arms (placebo/rosuvastatin) of missing IMT measurements (0, 1, 2 or 3 missing per IMT location) will be performed using a Chi-Square Test with a threshold of 1%.

#### 2. Analysis of the secondary endpoints:

To study rosuvastatin effect from baseline to week 48 on mean and / or of left and right maximal IMT progression, multi-levels, repeated measures, linear mixed-effects models adjusted for demographics and/or traditional CVD risk factors and centre will be used. Levels used for the data will be patient and carotid artery locations (CCA, ICA, BIF and ECA) within patients; the repeated measure will be time (baseline and week 48).

Repeated measures linear mixed-effects models adjusted for demographics and/or traditional CVD risk factors and centre will be used to assess the association between the arms (placebo/rosuvastatin) and each of the following parameters at week 0, 12, 24, 48, 72 and 96. We will test the interaction term between the arms and time (Month 0, 6, 12 and 24) to determine whether the rate of progression of the following parameters differed between arms (rosuvastatin versus placebo): Fasting Total Cholesterol, low-density lipoprotein (LDL)-cholesterol, high-density lipoprotein (HDL)-cholesterol, triglycerides and glucose.

Biomarkers of inflammatory process (sCD14, sCD163, neopterin, S-VCAM-1, adiponectin, CCL2, inflammatory (CD16+) monocyte expression of CD38, CX3CR1 and CD11b) will be

analysed using the same kind of regression with the same adjustments as described above including (LDL)-cholesterol and (HDL)-cholesterol.

The rate of adverse effects (symptomatic and biochemical) from the safety report will be summarized using frequency and percentage.

All efficacy analyses will compare the randomised treatment groups on an intention to treat basis regardless of treatments received during the study, including all patients with data at randomisation and at least one follow-up visit. Primary endpoint analyses will use a last value-carried forward approach for any patients permanently lost to follow-up. Secondary endpoints analyses will only include available data.

Statistical analysis will be performed using STATA Release 12.0 or updated version (Stata Statistical Software: Release 12.0, Stata Corporation, and College Station, USA).

We plan to recruit 102 patients. Drop outs will not be replaced unless the number surpasses the attrition rate of 15%.

An interim analysis will be performed at 48 weeks. The final analysis at 96 weeks will be conducted when all patients will have completed the follow-up visits or have been permanently lost to follow-up, and the study database is signed off as checked and complete.

#### 18 Insurance and Finances

Insurance for the Melbourne site is set up by AH and applies only to the one site. Insurance for Swiss sites is set up by the University Hospitals of Geneva (HUG) to cover the damages that may occur within this trial. The insurance applies to all Swiss participating study sites.

Swiss sites: Costs for the local laboratory tests (haematology, biochemistry, virology) that are not included in the routine HIV patient care will be covered by the patient care payments made to the sites by the leading site, Geneva.

# 19 Quality Control and quality assurance

#### 19.1 Source documents

Considered source documents are the patient's medical records including, but not limited to written electronic, magnetic and optical records and scans, x-rays, IMT images and electrocardiograms.

The following data will be considered source data:

- CRF: Compliance assessment, physical examination including measurements, smoking status, self-reported pregnancy or breast-feeding status
- Study medication distribution and return details.

## 19.2 Retention of essential documents

Essential documents as defined by ICH GCP include the signed protocol and any amendment(s), copies of the completed CRFs, signed Informed Consent Forms from all subjects who consented, hospital records, diary cards and other source documents, IRB/IEC
approvals and all related correspondence including approved documents, drug accountability records, trial correspondence and a list of the subject's names and addresses.

The Investigator must maintain all essential study documentation, and take measures to prevent accidental or premature destruction of these documents. The Investigator must retain the study documentation until at least ten years after completion or discontinuation of the study. After that period of time, the documents may be destroyed according local regulations.

#### 19.3 Data protection

Intima carotid ultrasound images will be coded with the subject's ID numbers and transferred for analysis to the cIMT Core Facility, Department of Medicine, **Montreal** Heart Institute, Université de Montréal, **Montreal**, Quebec, Canada **Responsible**: Pr Jean-Claude Tardif. Transfer of this data will be performed strictly anonymously (without personal identifiers), maintaining confidentiality and in line with both the Australian Privacy Law and the Swiss Federal Law on data protection that correspond to applicable laws of the province of Quebec, Canada.

Plasma samples will be coded with the subject's ID number and stored at the Burnet Institute 85 Commercial Rd, Melbourne, Victoria 3004 Australia or at the "sérothèque" (biobank) HUG in Switzerland. Swiss sites will ship the plasma samples to the central biobank ("sérothèque") of the HUG, 4, rue Gabrielle-Perret-Gentil 4, Geneva University Hospitals, Switzerland.

Samples may need to be transferred from Melbourne to Geneva or vice versa for analysis purposes. Shipment of plasma samples between the AH between AH (Burnet Institute, 85 Commercial Rd, Melbourne, Victoria 3004 Australia) and the HUG (Cardiology Laboratory, Hôpitaux Universitaires de Genève, Rue Gabrielle-Perret-Gentil 4, 1211 Geneva, Switzerland) for storage and testing of inflammatory markers will be performed strictly anonymously and in compliance with the Swiss Federal Law on data protection, which corresponds to applicable privacy laws of Australia and the state of Victoria, Melbourne.

#### 19.4 Monitoring, audits and inspections

Independent monitoring of the Swiss sites will be performed to ensure the strict implementation of the protocol and guidelines as well as to check consistency between the source data and the CRF in at least 50 percent of the number of enrolled subjects.

In case of audits or inspections by regulatory authorities or the ethics committee, the investigator will provide direct access to the original data, study documents and the sites facilities as well as to the site's personnel involved directly or indirectly in the trial.

### 20 Publications and presentations

The final data will be presented at one or more scientific meetings. No patient data will be presented that could permit identification of any individual study participant. Publication of data derived from this protocol will be supervised by the Principal Investigator in Melbourne and Geneva in conjunction with all study investigators. No other publication will be made before the primary manuscript has been agreed upon and accepted for publication and without prior approval of the principal investigator in Melbourne.

#### 21 References

- 1. D'Agostino RB, Sr., Vasan RS, Pencina MJ, et al. General cardiovascular risk profile for use in primary care: the Framingham Heart Study. Circulation 2008;117:743-53.
- 2. National Vascular Disease Prevention Alliance. Guidelines for the management of absolute cardiovascular disease risk. 2012. Accessed at www.heartfoundation.com.au
- 3. d'Arminio Monforte A, Sabin CA, Phillips A, et al. The changing incidence of AIDS events in patients receiving highly active antiretroviral therapy. Arch Intern Med 2005;165:416-23.
- 4. Palella FJ, Jr., Delaney KM, Moorman AC, et al. Declining morbidity and mortality among patients with advanced human immunodeficiency virus infection. HIV Outpatient Study Investigators. N Engl J Med 1998;338:853-60.
- 5. Obel N, Thomsen HF, Kronborg G, et al. Ischemic heart disease in HIV-infected and HIV-uninfected individuals: a population-based cohort study. Clin Infect Dis 2007;44:1625-31.
- 6. Lohse N, Hansen AB, Pedersen G, et al. Survival of persons with and without HIV infection in Denmark, 1995-2005. Ann Intern Med 2007;146:87-95.
- 7. Trevillyan J CA, Hoy J. Predictors of Coronary Heart Disease in HIV Positive Patients. 22nd Annual Conference of the Australasian Society for HIV Medicine 2010.
- 8. Bradshaw PJ, Alfonso HS, Finn J, Owen J, Thompson PL. A comparison of coronary heart disease event rates among urban Australian Aboriginal people and a matched non-Aboriginal population. J Epidemiol Community Health 2011;65:315-9.
- 9. Rose H, Hoy J, Woolley I, et al. HIV infection and high density lipoprotein metabolism. Atherosclerosis 2008;199:79-86.
- 10. Kuller LH, Tracy R, Belloso W, et al. Inflammatory and coagulation biomarkers and mortality in patients with HIV infection. PLoS Med 2008;5:e203.
- 11. Solages A, Vita JA, Thornton DJ, et al. Endothelial function in HIV-infected persons. Clin Infect Dis 2006;42:1325-32.
- 12. Parra S, Coll B, Aragones G, et al. Nonconcordance between subclinical atherosclerosis and the calculated Framingham risk score in HIV-infected patients: relationships with serum markers of oxidation and inflammation. HIV Med 2010;11:225-31.
- 13. Friis-Moller N, Sabin CA, Weber R, et al. Combination antiretroviral therapy and the risk of myocardial infarction. N Engl J Med 2003;349:1993-2003.
- 14. Friis-Moller N, Reiss P, Sabin CA, et al. Class of antiretroviral drugs and the risk of myocardial infarction. N Engl J Med 2007;356:1723-35.
- 15. Worm SW, Sabin C, Weber R, et al. Risk of myocardial infarction in patients with HIV infection exposed to specific individual antiretroviral drugs from the 3 major drug classes: the data collection on adverse events of anti-HIV drugs (D:A:D) study. J Infect Dis 2010;201:318-30.
- 16. Neuhaus J, Jacobs DR, Jr., Baker JV, et al. Markers of inflammation, coagulation, and renal function are elevated in adults with HIV infection. J Infect Dis 2010;201:1788-95.
- 17. Emery S, Neuhaus JA, Phillips AN, et al. Major clinical outcomes in antiretroviral therapy (ART)-naive participants and in those not receiving ART at baseline in the SMART study. J Infect Dis 2008;197:1133-44.
- 18. Kaplan RC, Sinclair E, Landay AL, et al. T cell activation and senescence predict subclinical carotid artery disease in HIV-infected women. J Infect Dis 2011;203:452-63.
- 19. Brenchley JM, Price DA, Schacker TW, et al. Microbial translocation is a cause of systemic immune activation in chronic HIV infection. Nat Med 2006;12:1365-71.
- 20. Ballou SP, Lozanski G. Induction of inflammatory cytokine release from cultured human monocytes by C-reactive protein. Cytokine 1992;4:361-8.

21. Chambless LE, Heiss G, Folsom AR, et al. Association of coronary heart disease incidence with carotid arterial wall thickness and major risk factors: the Atherosclerosis Risk in Communities (ARIC) Study, 1987-1993. Am J Epidemiol 1997;146:483-94.

Version 2.2

- 22. Bots ML, Palmer MK, Dogan S, et al. Intensive lipid lowering may reduce progression of carotid atherosclerosis within 12 months of treatment: the METEOR study. Journal of Internal Medicine 2009;265:698-707.
- 23. Hsue PY, Giri K, Erickson S, et al. Clinical features of acute coronary syndromes in patients with human immunodeficiency virus infection. Circulation 2004;109:316-9.
- 24. van Vonderen MGA, Hassink EAM, van Agtmael MA, et al. Increase in carotid artery intima-media thickness and arterial stiffness but improvement in several markers of endothelial function after initiation of antiretroviral therapy. Journal of Infectious Diseases 2009;199:1186-94.
- 25. van Vonderen MGA, Smulders YM, Stehouwer CDA, et al. Carotid intima-media thickness and arterial stiffness in HIV-infected patients: the role of HIV, antiretroviral therapy, and lipodystrophy. Journal of Acquired Immune Deficiency Syndromes: JAIDS 2009;50:153-61.
- 26. Duprez DA, Cohn JN. Arterial stiffness as a risk factor for coronary atherosclerosis. Curr Atheroscler Rep 2007;9:139-44.
- 27. Schillaci G, De Socio GVL, Pucci G, et al. Aortic stiffness in untreated adult patients with human immunodeficiency virus infection. Hypertension 2008;52:308-13.
- 28. van Wijk JPH, de Koning EJP, Cabezas MC, et al. Functional and structural markers of atherosclerosis in human immunodeficiency virus-infected patients. Journal of the American College of Cardiology 2006;47:1117-23.
- 29. Pirro M, Schillaci G, Mannarino MR, et al. Effects of rosuvastatin on 3-nitrotyrosine and aortic stiffness in hypercholesterolemia. Nutr Metab Cardiovasc Dis 2007;17:436-41.
- 30. Amarenco P, Labreuche J, Lavallee P, Touboul PJ. Statins in stroke prevention and carotid atherosclerosis: systematic review and up-to-date meta-analysis. Stroke 2004;35:2902-9.
- 31. Ridker PM, Danielson E, Fonseca FA, et al. Rosuvastatin to prevent vascular events in men and women with elevated C-reactive protein. N Engl J Med 2008;359:2195-207.
- 32. Ridker PM, Rifai N, Rose L, Buring JE, Cook NR. Comparison of C-reactive protein and low-density lipoprotein cholesterol levels in the prediction of first cardiovascular events. N Engl J Med 2002;347:1557-65.
- 33. Ridker PM, Cannon CP, Morrow D, et al. C-reactive protein levels and outcomes after statin therapy. N Engl J Med 2005;352:20-8.
- 34. Ridker PM, MacFadyen J, Libby P, Glynn RJ. Relation of baseline high-sensitivity C-reactive protein level to cardiovascular outcomes with rosuvastatin in the Justification for Use of statins in Prevention: an Intervention Trial Evaluating Rosuvastatin (JUPITER). American Journal of Cardiology 2010;106:204-9.
- 35. Jain MK, Ridker PM. Anti-inflammatory effects of statins: clinical evidence and basic mechanisms. Nat Rev Drug Discov 2005;4:977-87.
- 36. Mira E, Leon B, Barber DF, et al. Statins induce regulatory T cell recruitment via a CCL1 dependent pathway. J Immunol 2008;181:3524-34.
- 37. Montecucco F, Mach F. Update on statin-mediated anti-inflammatory activities in atherosclerosis. Semin Immunopathol 2009;31:127-42.
- 38. Dimitrow PP, Jawien M. Anti-inflammatory effect of atorvastatin in patients with aortic sclerosis or mild aortic stenosis independent of hypercholesterolemia. Pharmacol Rep 2010;62:1250-4.

- 39. Lewandowski M, Kornacewicz-Jach Z, Millo B, et al. The influence of low dose atorvastatin on inflammatory marker levels in patients with acute coronary syndrome and its potential clinical value. Cardiol J 2008;15:357-64.
- 40. Aslangul E, Fellahi S, Assoumou LK, Bastard JP, Capeau J, Costagliola D. Highsensitivity C-reactive protein levels fall during statin therapy in HIV-infected patients receiving ritonavir-boosted protease inhibitors. Aids 2011;25:1128-31.
- 41. Ganesan A, Crum-Cianflone NF, Higgins J, et al. High dose atorvastatindecreases cellular markers of immune activation: Results of a double-blind randomized controlled clinical trial. Journal of Infectious Diseases 2011;203:756-64.
- 42. Busti AJ, Bain AM, Hall RG, 2nd, et al. Effects of atazanavir/ritonavir or fosamprenavir/ritonavir on the pharmacokinetics of rosuvastatin. Journal of Cardiovascular Pharmacology 2008;51:605-10.
- 43. Kiser JJ, Gerber JG, Predhomme JA, Wolfe P, Flynn DM, Hoody DW. Drug/Drug interaction between lopinavir/ritonavir and rosuvastatin in healthy volunteers. J Acquir Immune Defic Syndr 2008;47:570-8.
- 44. Ageing AG-DoHa. General statement for lipid-lowering drugs prescribed as pharmaceutical benefits. In.
- 45. Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron 1976;16:31-41.
- 46. Kazmin A, Garcia-Bournissen F, Koren G. Risks of statin use during pregnancy: a systematic review. J Obstet Gynaecol Can 2007;29:906-8.
- 47. Walsh JC, Mandalia S, Gazzard BG. Responses to a 1 month self-report on adherence to antiretroviral therapy are consistent with electronic data and virological treatment outcome. Aids 2002;16:269-77.
- 48. The IDF consensus worldwide definition of the metabolic syndrome. (Accessed 20th April, 2012, at http://www.idf.org/webdata/doc/IDF Meta def final.pdf.)
- 49. Thygesen K, Alpert JS, White HD. Universal definition of myocardial infarction. Eur Heart J 2007;28:2525-38.
- 50. Friis-Moller N, Thiebaut R, Reiss P, et al. Predicting the risk of cardiovascular disease in HIV-infected patients: the data collection on adverse effects of anti-HIV drugs study. Eur J Cardiovasc Prev Rehabil 2010;17:491-501.
- 51. Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med 1999;130:461-70.

### 22 Appendix

### **22.1 Case Record Forms**

### 22.1.1 Screening Visit

| Screening Visit – Rosuvastatin Trial | |
|---|---|
| Screening Number | |
| Date | |
| Informed Consent Signed | □ Yes □ No |
| Age (years – round number) | |
| Gender | ☐ Male ☐ Female |
| Ethnicity | ☐ Caucasian |
| | ☐ Asian |
| | ☐ African |
| | ☐ Aboriginal/Torres Strait Islander |
| Date first diagnosed with HIV | |
| <b>Prior AIDS defining illnesses</b> | □ Yes □ No |
| List any previous AIDS defining illness | 1. |
| | 2. |
| | 3. |
| | 4. |
| | 5. |
| | 6. |
| | 7. |
| Currently taking antiretrovirals | □ Yes □ No |
| Change in antiretroviral in last six (6) | □ Yes □ No |
| Total cumulative years on Indinavir | |
| Total cumulative years on lopinavir | |
| HIV Viral load been <200 copies/ml for | □ Yes □ No |
| CD4+ T-cell Nadir | |
| List all past medical history | 1. |
| (Tick box if currently active/being treated) | 2. |
| (Tick box if currently active/being freated) | 3. |
| | 4. |
| | 5. |
| | 6. |
| | 7. |
| | 8. |
| | 9. |

| | 10. |
|----------------------------------------------|------------------|
| | 11. |
| | 12. |
| Specifically ever diagnosed with: | - |
| a. Coronary Heart Disease/AMI | □ Yes □ No |
| b. Angina | □ Yes □ No |
| c. Diabetes | □ Yes □ No |
| d. Stroke | □ Yes □ No |
| e. Transient Ischaemic attack | □ Yes □ No |
| f. Peripheral vascular disease | □ Yes □ No |
| g. Hypertension | □ Yes □ No |
| h. Hypercholesterolemia | □ Yes □ No |
| i. Familial Hypercholesterolemia | □ Yes □ No |
| j. Myopathy | □ Yes □ No |
| Exposure to the following drugs in last | |
| a. Statins | □ Yes □ No |
| b. Ezetimibe | □ Yes □ No |
| c. Fibrates | □ Yes □ No |
| d. Niacin | □ Yes □ No |
| e. Anti-hypertensives | □ Yes □ No |
| f. Anti-platelets | □ Yes □ No |
| Pregnant? | □ Yes □ No |
| Breast Feeding? | □ Yes □ No |
| Smoking status | ☐ Never Smoked |
| | ☐ Ex-smoker |
| | ☐ Current smoker |
| IF ex-smoker: | |
| Time since quitting | |
| Estimated quantity/day when was smoking | |
| Duration of smoking history (years) | |
| IF current smoker | |
| Estimated quantity/day | |
| Duration of smoking history (years) | |
| Family history of heart disease | □ Yes □ No |
| Age of Diagnosis in male 1st degree relative | |
| Age of Diagnosis in female 1st degree | |

| | <b>Current Antiretroviral Med</b> | dications | |
|---|---|---|---|
| Trade Name | Generic Name | Daily Dose | Start Date |
| 1. | | | |
| 2. | | | |
| 3. | | | |
| 4. | | | |
| 5. | | | |
| 6. | | | |
| C | Concomitant Medications / Su | upplements | |
| Trade Name | Generic Name | Daily Dose | Start Date |
| 1. | | | |
| 2. | | | |
| 3. | | | |
| 4. | | | |
| 5. | | | |
| 6. | | | |
| 7. | | | |
| 8. | | | |
| 9. | | | |
| 10. | | | |
| 11. | | | |
| 12. | | | |
| 13. | | | |
| 14. | | | |
| 15. | | | |
| 16. | N/ 11 / All 1 | | |
| NI CNT I' ' | Medication Allergie | | |
| Name of Medicatio | on Des | scription of allergy | / |
| 1. | | | |
| 2. 3. | | | |
| 4. | | | |
| 5. | | | |
| J. | | | |

| Examination | | | | |
|---------------------------------------|---------|----|----|--------|
| Height (m) | | | | |
| Weight (kg) | | | | |
| Waist circumference (cm) | | | | |
| Peripheral pulses | □ prese | nt | | absent |
| Systolic Blood Pressure | | | | |
| Diastolic Blood Pressure | | | | |
| Physical examination | | | | |
| (Document any relevant abnormalities) | | | | |
| Date ECG performed | | | | |
| Date cIMT performed | | | | |
| Date cPWV performed | | | | |
| Date bloods taken | | | | |
| Once Results available: | | | | |
| Creatinine clearance | | | | |
| Framingham Risk score | | | | |
| Is patient eligible for enrolment | □ Yes | | No | |
| If No, please document why | | | | |
| If yes, Randomisation number | | | | |

## **Inclusion / Exclusion Checklist**

| INCLUSION CRITERIA | | | |
|---|---|---|---|
| Signed consent form | | YES | □ NO |
| Age ≥ 30 years | | YES | ☐ NO |
| Framingham Risk Score of 10-15% [FRS =] | | YES | ☐ NO |
| HIV positive | | YES | ☐ NO |
| Stable cART regimen for ≥ 6 months | | <b>YES</b> | ☐ NO |
| HIV viral load <200copies/ml for ≥ 6 months | | <b>YES</b> | NO |
| EXCLUSION CRITERIA | | | |
| | | YES | □NO |
| Coronary heart disease (CHD), stroke or PVD | | | |
| Family history of CHD < 55 in a male <u>first</u> degree relat | ive | YES | ∐ NO |
| Family history of CHD <65 in a female <u>first</u> degree relative | | YES | NO |
| Type 2 Diabetes | | YES | ☐ NO |
| Familial hypercholesterolaemia | | <b>YES</b> | ☐ NO |
| Aboriginal or Torres Strait Islander people with LDL-C >2.5 mmol/L | | YES | □ NO |
| Blood pressure ≥ 180/110 | | YES | ☐ NO |
| HDL-C < 1 mmol/L and total cholesterol > 6.5 mmol/L | | YES | □ NO |
| Documented history of: | | | |
| Ischemic stroke or transient ischemic attack (TIA) | | YES | □ NO |
| Peripheral arterial disease (regardless of severity) | | YES | ☐ NO |
| Congestive heart failure | | YES | ☐ NO |
| Coronary artery disease or ECG findings consistent with prior MI | h | YES | □ NO |
| Carotid artery stenosis or >50% occlusion of carotid | | | |
| artery known previously or discovered during screeni | ing | YES | ☐ NO |
| procedures | | | |
| Total cholesterol >7.5 mmol/L | | YES | □ NO |

| Triglyceride level > 4 mmol/L | | YES | □ NO |
|---|---|---|---|
| HDL-c <1mmol/l and total cholesterol >6.5mmol/l | | YES | NO |
| Current or prior (last 6 months) statin therapy | | YES | □ NO |
| Current or prior (last 6 months) use of ezetimibe | | YES | □ NO |
| Current or prior (last 6 months) use of fibrates or niacin | | YES | □ NO |
| Pregnancy or lactation | | <b>YES</b> | ☐ NO |
| Hypersensitivity to statins | | <b>YES</b> | ☐ NO |
| Known myopathy or baseline CK > 3x ULN | | <b>YES</b> | ☐ NO |
| Contraindicated concurrent medication (to statin use) | | YES | ☐ NO |
| Current cyclosporine, fusidic acid or oral corticosteroid use | | YES | NO |
| Concomitant antiplatelet drug | | YES | ☐ NO |
| Unable to complete study procedures (i.e. attendance at AH for cIMT and cPWV testing or cIMT images not accepted for analysis despite redo examination) | | YES | □ NO |
| Conocmitant renal or hepatic disease, defind as the presence of the following: | YES | □ NO | |
| Creatinine clearance <30 ml/min [CCL =] | YES | □ NO | |
| Transaminases (ALT, AST) >3x the upper limit of normal | YES | □ NO | |
| Acute hepatic failure | YES | ☐ NO | |
| Compensated cirrhosis Child Class B or C | YES | ☐ NO | |
| Other active significant disease | YES | ☐ NO | |
| - Describe | | | |
| Eligible for Trial? | YES | □ NO | |
| Completed by: | | | |
| Signed | Date / | / | |

### 22.1.2 Baseline Visit

| Study number | | | | |
|---|---|---|---|---|
| Date of Visit | | / | / | |
| Any new medical diagnosis | since | □ Yes | □ No | |
| screening? | | 1. | | |
| If yes, list: | | 2. | | |
| | | 3. | | |
| | | 4. | | |
| Any new medications since l | last visit? | □ Yes | □ No | |
| If yes please detail below | | | | |
| Trade Name | Gene | eric Name | Daily Dose | Start Date |
| 1. | | | | |
| 2. | | | | |
| 3. | | | | |
| Any medications ceased since last visit? If yes please detail below | | □ Yes | □ No | |
| Trade Name | Gen | eric Name | Daily Dose | Stop Date |
| 1. | | | | |
| 2. | | | | |
| 3. | | | | |
| Smoking status | | □ Non-smo | oker | |
| | | ☐ Ex- Smoker | | |
| | | ☐ Current smoker | | |
| Has an adverse event occurr | red? | □ Yes □ No | | |
| If yes please complete adver | se event | | | |
| Any new abnormalities on | | ☐ Yes ☐ No | | |
| If yes list: | | 1. | | |
| | | 2. | | |
| | | 3. | | |
| Weight (kg) | | | | |
| <b>Blood Pressure</b> | | | | |
| Provided with 3/12 supply of | | □ Yes | □ No | |
| Bloods taken? | | □ Yes | □ No | |
| Commission by | | C: | | |
| Completed by: | | Signed | | |

### 22.1.3 Week 12 Visit

| Study number | | | | |
|---|---|---|---|---|
| Date of Visit | | / | <u>/</u> | |
| Any new medical diagnosis | since | □ Yes | □ No | |
| screening? | | 1. | | |
| If yes, list: | | 2. | | |
| | | 3. | | |
| | | 4. | | |
| Any new medications since l | ast visit? | □ Yes | □ No | |
| If yes please detail below | | | | |
| Trade Name | Gene | eric Name | Daily Dose | Start Date |
| 1. | | | | |
| 2. | | | | |
| 3. | | | | |
| Any medications ceased sinc | re last | □ Yes | □ No | |
| visit? If yes please detail bel | | | | |
| Trade Name | Gene | eric Name | Daily Dose | Stop Date |
| 1. | | | | |
| 2. | | | | |
| 3. | | | | |
| Smoking status | | □ Non-smo | ker | |
| | | ☐ Ex- Smoker | | |
| | | ☐ Current smoker | | |
| Has an adverse event occurr | red? | □ Yes □ No | | |
| Myopathic symptoms | | □ Yes □ No | | |
| Gastrointestinal disturbance | e | □ Yes | □ No | |
| Jaundice | | □ Yes | □ No | |
| If yes please complete adver | se event | | | |
| Any new abnormalities on | | □ Yes | □ No | |
| If yes list: | | 1. | | |
| | | 2. | | |
| | | 3. | | |
| Weight (kg) | | | | |
| <b>Blood Pressure</b> | | | | |
| Bloods taken? | | □ Yes | □ No | |
| Completed by: | | Signed | | |

### **22.1.4** Week 24 Visit

| Study number | | | | |
|---|---|---|---|---|
| Date of Visit | Date of Visit | | / | |
| Any new medical diagnosis | since | □ Yes □ No | | |
| screening? If yes, list: | | 1. | | |
| | | 2. | | |
| | | 3. | | |
| | | 4. | | |
| Any new medications since | last visit? | □ Yes | □ No | |
| If yes please detail below | | | | |
| Trade Name | Gene | eric Name | Daily Dose | Start Date |
| 1. | | | | |
| 2. | | | | |
| 3. | | | | |
| Any medications ceased since | ce last | □ Yes | □ No | • |
| visit? If yes please detail bel | | | | |
| Trade Name | Gene | eric Name | Daily Dose | <b>Stop Date</b> |
| 1. | | | | |
| 2. | | | | |
| 3. | | | | |
| <b>Smoking status</b> | • | □ Non-sn | noker | • |
| | | ☐ Ex-Sm | oker | |
| | | ☐ Current smoker | | |
| Has an adverse event occurr | red? | □ Yes □ No | | |
| Myopathic symptoms | | □ Yes □ No | | |
| Gastrointestinal disturbance | e | □ Yes | □ No | |
| Jaundice | | □ Yes | □ No | |
| If yes please complete adver | se event | | | |
| Any new abnormalities on | | □ Yes | □ No | |
| If yes list: | | 1. | | |
| | | 3. | | |
| Weight (kg) | | | | |
| <b>Blood Pressure</b> | | | | |
| Bloods taken? | | □ Yes | □ No | |
| Completed by: | | Signed | | |

| 22.1.5 Week 48 Visit | | | | |
|---|---|---|---|---|
| Study number | | | | |
| Date of Visit | | / | / | |
| Any new medical diagnosis since screening? | | □ Yes | □ No | |
| | | 1. | | |
| If yes, list: | | 2. | | |
| | | 3. | | |
| | | 4. | | |
| Any new medications since l | last visit? | □ Yes | □ No | |
| If yes please detail below | | | | |
| Trade Name | Gen | eric Name | Daily Dose | Start Date |
| 1. | | | | |
| 2. | | | | |
| 3. | | | | |
| Any medications ceased since | re last | □ Yes | | |
| visit? If yes please detail be | | | | |
| Trade Name | | eric Name | Daily Dose | <b>Stop Date</b> |
| 1. | | | | |
| 2. | | | | |
| 3. | | | | |
| Smoking status | | □ Non-sn | ıoker | |
| | | ☐ Ex- Smoker | | |
| | | ☐ Current smoker | | |
| Has an adverse event occurr | red? | ☐ Yes ☐ No | | |
| Myopathic symptoms | | □ Yes | □ No | |
| Gastrointestinal disturbance | e | □ Yes | □ No | |
| Jaundice | | □ Yes | □ No | |
| If yes please complete adver | se event | | | |
| Any new abnormalities on | | □ Yes | □ No | |
| If yes list: | | 1. | | |
| | | 2. | | |
| | | 3. | | |
| Weight (kg) | | | | |
| Blood Pressure | | | | |
| Compliance assessment per | formed | □ Yes | □ No | |
| Bloods taken? | | | | |
| Date cIMT/PWV performed | l /booked | | | |
| Completed by: | | Signed | | |

#### **Compliance Assessment Week 48 study Visit**

| Study Numb | er | <br> |
|------------|----|------|
| Date/ | ·/ | |

We understand that many people on medications find it very difficult to take them regularly, and often miss doses. It is important for us to know how many doses of the study medication you've missed.

Version 2.2

<u>This questionnaire is completely confidential</u>. Your answers will not be shown to your doctor or others involved in your care

How many doses (tablets) have you missed in the last seven (7) days?

How many doses (tablets) have you missed in the last **twenty-eight (28)** days?

Put an X on the line below at the point showing <u>your best guess</u> about how much of the study medication you have taken *during the past 28 days*.

For example, 0% means you haven't taken any dose of the medication above, 50% means you have taken half of the prescribed doses of the medication above and 100% means you have taken every single dose of the medication above



### 22.1.6 Week 72 Visit

| Study number | | | | |
|---|---|---|---|---|
| Date of Visit | | / | / | |
| Any new medical diagnosis s | since | □ Yes | □ No | |
| screening? | | 1. | | |
| If yes, list: | | 2. | | |
| | | 3. | | |
| | | 4. | | |
| Any new medications since l | ast visit? | □ Yes | □ No | |
| If yes please detail below | | | | |
| Trade Name | Gene | eric Name | Daily Dose | Start Date |
| 1. | | | | |
| 2. | | | | |
| 3. | | | | |
| Any medications ceased sinc | e last | □ Yes | □ No | |
| visit? If yes please detail belo | OW | | | |
| Trade Name | Gene | eric Name | Daily Dose | Stop Date |
| 1. | | | | |
| 2. | | | | |
| 3. | | | | |
| Smoking status | | □ Non-smol | ker | |
| | | ☐ Ex-Smoker | | |
| | | ☐ Current s | smoker | |
| Has an adverse event occurr | ed? | □ Yes □ No | | |
| Myopathic symptoms | | □ Yes □ No | | |
| Gastrointestinal disturbance | <u>)</u> | □ Yes □ No | | |
| Jaundice | | □ Yes | □ No | |
| If yes please complete advers | se event | | | |
| Any new abnormalities on | | □ Yes | □ No | |
| If yes list: | | 1. | | |
| | | 2. | | |
| | | 3. | | |
| Weight (kg) | | | | |
| <b>Blood Pressure</b> | | | | |
| Bloods taken? | | □ Yes | □ No | |

| Completed by: | Signed |
|---------------|--------|
| = | |

### 22.1.7 Week 96 Visit

| Study number | | | | |
|---|---|---|---|---|
| Date of Visit | | / | | |
| Any new medical diagnosis since | | □ Yes □ No | | |
| screening? | | 1. | | |
| If yes, list: | | 2. | | |
| | | 3. | | |
| | | 4. | | |
| Any new medications since l | ast visit? | □ Yes | □ No | |
| If yes please detail below | | | | |
| Trade Name | Gene | ric Name | Daily Dose | Start Date |
| 1. | | | | |
| 2. | | | | |
| 3. | | | | |
| Any medications ceased sinc | e last | □ Yes | □ No | |
| visit? If yes please detail belo | OW | | | |
| Trade Name | Gene | ric Name | Daily Dose | Stop Date |
| 1. | | | | |
| 2. | | | | |
| 3. | | | | |
| Smoking status | | Non-smoker | | |
| (circle whichever is appropr | iate) | Ex- Smoker | | |
| | | Current smoker | | |
| Has an adverse event occurr | ed? | □ Yes | □ No | |
| Myopathic symptoms | | □ Yes □ No | | |
| Gastrointestinal disturbance | | □ Yes | □ No | |
| Jaundice | | □ Yes | □ No | |
| If yes please complete advers | se event | | | |
| Any new abnormalities on | | □ Yes | □ No | |
| If yes list: | | 1. | | |
| | | 2. | | |
| | | 3. | | |
| Weight (kg) | | | | |
| <b>Blood Pressure</b> | | | | |
| Compliance assessment performed | | □ Yes | □ No | |
| Bloods taken? | | | | |
| Date cIMT/PWV performed | /booked | | | |
| | | - | | |

Completed by: \_\_\_\_\_Signed \_\_\_\_

#### **Compliance Assessment Week 96 study Visit**

| <b>Study Numb</b> | er |
|-------------------|----|
| Date | // |

We understand that many people on medications find it very difficult to take them regularly, and often miss doses. It is important for us to know how many doses of the study medication you've missed.

<u>This questionnaire is completely confidential</u>. Your answers will not be shown to your doctor or others involved in your care

How many doses (tablets) have you missed in the last seven (7) days?

How many doses (tablets) have you missed in the last **twenty-eight (28)** days?

Put an X on the line below at the point showing <u>your best guess</u> about how much of the study medication you have taken *during the past 28 days*.

For example, 0% means you haven't taken any dose of the medication above, 50% means you have taken half of the prescribed doses of the medication above and 100% means you have taken every single dose of the medication above



### **22.1.8 Unscheduled Visits**

| Study Number | |
|---|---|
| Date of Visit | /Time::hr |
| Person initiating unscheduled | |
| Reason for unscheduled visit | |
| <b>Adverse Event Assessment</b> | |
| Onset date of Adverse Event | |
| Time of Onset (if Known) | |
| <b>Description of Adverse event:</b> | |
| <b>Adverse Event Severity Grade</b> | ☐ Mild (Grade 1) |
| (refer to Division of AIDS Table | ☐ Moderate (Grade 2) |
| for grading of severity) | ☐ Severe (grade 3-4) |
| Is this a Serious Adverse Event | $\square$ Yes $\square$ No (If YES, please fill in the |
| Treatment for AE required? | □ Yes □ No |
| (If yes describe in detail) | |
| Related to the study drug? | ☐ Confirmed |
| | ☐ Probable |
| | ☐ Possible |
| | ☐ Excluded |
| | ☐ Non -assessable |
| Study medication stopped | □ Yes □ No |
| Withdrawn from the study | □ Yes □ No |
| <b>Outcome of Adverse Event</b> | □ Ongoing |
| | ☐ Resolved |
| | □ Unknown |
| Date of resolution of adverse | /(If not ongoing) |
| Date subject will be next | |
| Completed by: | Signed |

22.2 Serious Adverse Event (SAE) Form

| Study Number | |
|----------------------------------|-----------------------------------------|
| Date of Awareness | /TIME::h |
| Onset Date of Event | /TIME::h |
| Stop Date of Event | /TIME::h |
| Type of Report | ☐ Initial ☐ Follow-up ☐ Final |
| Description of SAE: | |
| Category of SAE | ☐ Death Date of Death/ |
| | ☐ Life Threatening |
| | ☐ Caused or prolonged hospitalization |
| | ☐ Resulted in significant disability or |
| | ☐ Other important medical condition |
| Related to the study drug? | ☐ Confirmed |
| | ☐ Probable |
| | ☐ Possible |
| | ☐ Excluded |
| | □ Non -assessable |
| If Adverse Drug reaction please | |
| - Generic name | |
| - Lot Number | |
| - Dosage | |
| - Route of administration | |
| - Start date | / |
| - Indication | |
| Study medication stopped? | □ Yes □ No |
| If yes did the AE resolve after | □ Yes □ No |
| Was the code broken? | □ Yes □ No |
| If YES, what was the allocation? | |
| Treatment for SAE required? | □ Yes □ No |
| (If yes describe in detail) | |
| Completed by:Signo | ed Date/ |

### 22.3 Units of measurement and reference ranges

| Investigation | Abbreviation | Units | Reference Range |
|---|---|---|---|
| HIV specific tests | | | |
| CD4+ T-cell count | - | cells/μL | 410 - 1,545 |
| HIV Viral Load | - | copies/ml | < 20 |
| Full Blood Examination (FBE) | Full Blood Examination (FBE) | | |
| Haemoglobin | Hb | g/L | 128 - 175 |
| Total White Cell count | WCC | cells x109/L | 3.9 – 12.70 |
| Lymphocytes | Lymp | cells x109/L | 0.9 – 3.30 |
| Neutrophils | Neut | cells x109/L | 1.9 – 8.0 |
| Platelets | Plt | cells x109/L | 150 - 396 |
| Biochemistry | | | |
| Sodium | Na | mmol/L | 135 – 143 |
| Potassium | K+ | mmol/L | 3.5 – 5.0 |
| Chloride | Cl | mmol/L | 99 - 107 |
| Bicarbonate | НСО3 | mmol/L | 20 - 32 |
| Calcium | Ca | mmol/L | 2.14 – 2.50 |
| Phosphate | PO <sub>4</sub> | mmol/L | 0.6 – 1.30 |
| Urea | Ur | mmol/L | 4.0 – 9.0 |
| Creatinine | Cr | μmol/L | 60 - 105 |
| Estimated glomerular filtration rate | eGFR | ml/min | > 90 |
| Beta Human chorionic gonadotrophin | βHCG | U/L | < 3 |
| High sensitivity C- reactive protein | hsCRP | mg/L | < 5.0 |
| Creatinine phosphokinase | СРК | U/L | 60 - 285 |
| Liver Function Tests (LFT) | | | |
| Total Protein | ТР | g/L | 60 - 80 |

| Albumin | Alb | g/L | 33 - 46 |
|---|---|---|---|
| Bilirubin | Bil | μmol/L | < 23 |
| Alanine Aminotransferase | ALT | U/L | 12-52 |
| Alkaline Phosphatase | ALP | U/L | 42 - 125 |
| Gamma- glutamyl transpeptidase | GGT | U/L | < 62 |
| Fasting Metabolic Assessments | | | |
| Total Cholesterol | TC | mmol/L | < 5.5 |
| High Density Lipoprotein Cholesterol | HDL-C | mmol/L | > 1.0 |
| Low Density Lipoprotein Cholesterol | LDL-C | mmol/L | < 3.5 |
| Triglycerides | TG | mmol/L | < 2.0 |
| Glucose | - | mmol/L | 3.8 – 7.7 |
| Structural / Physical Assessments | | | |
| Carotid intima media thickness | cIMT | mm | n/a |
| Carotid-femoral pulse wave velocity | cPWV | m/s | n/a |
| Height | - | Meters (m) | n/a |
| Weight | - | Kilograms<br>(Kg) | n/a |
| Calculations | | | |
| Body Mass Index | BMI | kg/m2 | <ul> <li>&lt; 18.5 Underweight</li> <li>18.5 - 24.9 Healthy</li> <li>25.0 - 29.9 Overweight</li> <li>30.0 - 34.9 Obesity I</li> <li>35.0 - 39.9 Obesity II</li> <li>&gt; 40 Obesity III</li> </ul> |
| Framingham Risk Score | FRS | % 10 year<br>risk | < 10 % Low Risk<br>10 -15 % Moderate Risk<br>> 15 % High risk |
| D.A.D. Risk Score | DRS | % 5 year risk | < 1% Low Risk 1 – 5% Moderate Risk 5 – 10% High Risk > 10% Very High Risk |
| Estimated creatinine clearance | CrCl | ml/min | > 90 |

### 22.4 Units of measurement and reference ranges for Swiss sites

| Investigation | Abbreviation | Units | Reference Range |
|---|---|---|---|
| HIV specific tests | | | |
| CD4+ T-cell count | - | cells/µl | 600 – 1'950 |
| HIV Viral Load | - | copies/ml | < 20 |
| Full Blood Examination (FBE) | Full Blood Examination (FBE) | | |
| Haemoglobin | НЬ | g/L | M: 140-180 F: 120-160 |
| Total White Cell count | WCC | G/L | 4.0 – 11.0 |
| Lymphocytes | Lymp | G/L | 1.00 - 4.50 |
| Neutrophils | Neut | G/L | 1.50-8.00 |
| Platelets | Plt | G/L | 150-350 |
| Biochemistry | | | |
| Sodium | Na | mmol/L | 136-144 |
| Potassium | K+ | mmol/L | 3.6 – 4.6 |
| Chloride | Cl | mmol/L | 96 - 107 |
| Bicarbonate | HCO <sub>3</sub> | mmol/L | 23.0-30.0 |
| Calcium | Ca | mmol/L | 2.20-2.52 |
| Phosphate | PO <sub>4</sub> | mmol/L | 0.8-1.5 |
| Urea | Ur | mmol/L | 2.8-7.1 |
| Creatinine | Cr | μmol/L | M: 62-106 F: 35-88 |
| Estimated glomerular filtration rate | eGFR | ml/min | > 90 |
| Beta Human chorionic gonadotrophin | β HCG | U/L | |
| Creatinine phosphokinase | СРК | U/L | M: 47-222 F:33-187 |
| Liver Function Tests (LFT) | | | |
| Total Protein | TP | g/L | 61-79 |
| Albumin | Alb | g/L | 35-48 |

| Bilirubin | Bil | μmol/L | 6.8-25 |
|---|---|---|---|
| Alanine Aminotransferase | ALT | U/L | M: 12 - 50 F: 9 - 42 |
| Alkaline Phosphatase | ALP | U/L | 30 - 125 |
| Gamma- glutamyl transpeptidase | GGT | U/L | M: 9 - 40 F: 9 - 35 |
| Fasting Metabolic Assessments | | | |
| Total Cholesterol | TC | mmol/L | < 6.5 |
| High Density Lipoprotein Cholesterol | HDL-C | mmol/L | M: >0.90 F: > 1.00 |
| Low Density Lipoprotein Cholesterol | LDL-C | mmol/L | < 4.0 |
| Triglycerides | TG | mmol/L | < 2.00 |
| Glucose | - | mmol/L | 4.1 – 6.0 |

#### 22.5 Patient Informed Consent Form



# Participant Information Sheet/Consent Form Interventional Study - Adult providing own consent

#### The Alfred Hospital

Title Does Rosuvastatin delay progression of

atherosclerosis in people with HIV infection? A multicentre randomized, double blind placebo-

controlled trial

Coordinating Principal Investigator/

**Principal Investigator** 

Dr Janine Trevillyan Prof Jennifer Hoy

Associate Investigator(s) Professor Suzanne Crowe

Dr Julian Elliott

A. Professor Anthony Jaworowski

Dr James Shaw

**Professor Anthony Dart** 

**Location** The Alfred Hospital

#### Part 1 What does my participation involve?

#### 1 Introduction

You are invited to take part in this research project. This is because you have human immunodeficiency virus (HIV) infection, are currently on anti-HIV medications and are thought to have a moderate risk of developing heart disease. The research project is testing a new treatment to prevent heart disease in HIV positive people. The new treatment is called Rosuvastatin, a cholesterol lowering medication.

This Participant Information Sheet/Consent Form tells you about the research project. It explains the tests and treatments involved. Knowing what is involved will help you decide if you want to take part in the research.

Please read this information carefully. Ask questions about anything that you don't understand or want to know more about. Before deciding whether or not to take part, you might want to talk about it with a relative, friend or your local doctor.

Participation in this research is voluntary. If you don't wish to take part, you don't have to. You will receive the best possible care whether or not you take part.

If you decide you want to take part in the research project, you will be asked to sign the consent section. By signing it you are telling us that you:

- Understand what you have read
- Consent to take part in the research project

- Consent to have the tests and treatments that are described
- Consent to the use of your personal and health information as described.

You will be given a copy of this Participant Information and Consent Form to keep.

#### 2 What is the purpose of this research?

Since people started taking anti-HIV medications, illness from AIDS has decreased, but other serious diseases like heart disease (heart attacks) and other diseases of blood vessels (such as strokes) have increased. HIV causes inflammation (irritation) inside the body that cannot be felt but can be measured by certain blood tests. Inflammation may contribute to diseases (such as heart attacks) by damaging blood vessels. HIV therapy can partially lower inflammation, however the levels of inflammation in people who have HIV may remain high even when they are on anti-HIV medications compared with those found in people who do not have HIV.

The main goal of this study is to see if taking rosuvastatin (a cholesterol lowering medication that also decreases inflammation) will slow down the development of blood vessel damage (a sign of future heart attacks) in people infected with HIV who are at moderate risk of heart disease and so are not currently eligible for rosuvastatin.

In addition to observing the effects of rosuvastatin on the level of inflammation measured in the blood, this study will see if rosuvastatin is safe for people with HIV who are also taking medication for HIV.

Medications, drugs and devices have to be approved for use by the Australian Federal Government. Rosuvastatin is approved in Australia to treat high cholesterol levels in the blood and to prevent heart attacks in people at high risk or who have already had a heart attack. However it has not been approved for use in patients who are at moderate risk. Therefore, it is an experimental treatment. This means that it must be tested to see if it is an effective therapy to prevent heart disease in people at moderate risk. Rosuvastatin has been able to lower the level of inflammation in certain other diseases but has not been studied for this purpose in people who have HIV.

The results of this research will be used by the study doctor, Dr Janine Trevillyan to obtain a PhD degree.

This research has been initiated by the study doctor, Professor Jennifer Hoy and is funded through Monash University.

#### 3 What does participation in this research involve?

If you choose to participate in this project you will be asked to sign this consent form prior to any study assessments being performed. If you would like an interpreter to be present at any time we will arrange one for you.

You will be participating in a randomised controlled research project. Sometimes we do not know whether a medication is going to prevent a particular condition. To find out we need to compare the treatment to having no treatment at all. We do this by putting people into groups and giving one group the treatment (Rosuvastatin) and one group a placebo. The results from each group are compared to see if one is better. A placebo is a medication with no active ingredients or any medical benefit. It looks like the real thing but is not. To try to make sure the groups are the same, each participant is put into a group by chance (random). You will have a 50/50 (equal) chance of being in either group.

You will need to take one capsule a day which will contain either the placebo or 20mg of rosuvastatin. Some HIV medications (in particular those from the group of drugs known as protease inhibitors) can cause the level of rosuvastatin to rise. If you are on one of these medications you will be given 10mg of rosuvastatin (or placebo) instead.

Version 2.2

You will be participating in a double-blind study. This means that neither you nor your study doctor will know which treatment you are receiving. However, in certain circumstances your study doctor can find out which treatment you are receiving.

This research project has been designed to make sure the researchers interpret the results in a fair and appropriate way and avoids study doctors or participants jumping to conclusions.

#### **Evaluations performed during the study**

If you decide to take part in the research project you will be asked some questions about your medical history, the medications you take and any risk factors you have that might predispose you to developing heart disease. We will check how well your liver is functioning and your cholesterol levels. This will let us know if you are eligible to take part. Completing the screening visit will take approximately 15- 30 minutes.

The study visits will occur at the same time as your routine HIV visits with your primary care doctor as far as is possible, and will take between 30 – 45 minutes depending on how many tests need to be performed. At the first visit and four times during the study you will be asked not to eat or drink anything (other than your required medications and normal amounts of plain water) for at least 8 hours (preferably 12 hours) before you come in for blood tests.

At the study visits you will be asked about your health and any medicines you have taken. You will be weighed and have your blood pressure checked and will be asked how often you have taken your medications over the few days and weeks prior to the visit.

At each study visit you will have blood tests taken to check for side effects of the medication and to monitor your liver function. Every six months there will also be blood taken to test for signs of inflammation, cholesterol levels, CD4 (T cell) counts and HIV viral loads.

Prior to starting the rosuvastatin or placebo and at 12 months and 24 months, (the end of the study), you will have an ultrasound of your carotid arteries (the large arteries in your neck) to measure the thickness of the artery wall (which allows us to estimate your chance of developing heart disease). This is a painless procedure that takes about 20 minutes. On the same day we will also measure the speed your blood flows to the carotid artery (in your neck) and the femoral artery (at the top of your thigh). This is done with a machine very similar to an ultrasound and is also painless. It takes about 10 minutes. Both of these tests are performed onsite at the Alfred Hospital.

If at any time during the study you develop a side effect from the medication you may need to come in for an extra visit to check on your safety. You will be assessed by the study doctor and advised whether you should stop the study medication and whether you require any other treatment or investigation.

You will be involved in this study for ninety-six (96) weeks, approximately 2 years. The study will run for five years in total and will be monitored by an independent review board.

There are no additional costs associated with participating in this research project, nor will you be paid. All medication, tests and medical care required as part of the research project will be provided to you free of charge.

You will have to pay for your usual medicines (including HIV medications) like you normally would.

#### 4 What do I have to do?

You do not need to change your diet or level of exercise to participate in this study.

You should keep taking your usual medications (including your HIV medications) throughout the study which will be guided by your usual HIV doctor. If you are taking warfarin your INR level will need to be monitored more often than usual when you first start taking the study drug.

You should not start any of the medications listed below while you're in this study because they may increase your chance of developing a side effect.

- Cholesterol lowering medications including niacin, fibrates or 'statins'
- Fusidic acid (an antibiotic)
- Cyclosporine

Please tell the study team if you need to start any new medications so that they can check if it will be safe to take while taking rosuvastatin.

You can still donate blood while in this study if you wish.

People who have had side effects from cholesterol lowering medications before or have significant problems with their liver or muscles cannot take part in this study. If you are pregnant or planning on becoming pregnant in the next two years you cannot take part in this study.

To be part of the study you need to commit to taking the study medication every day.

#### 5 Other relevant information about the research project

102 people will be taking part in the project. Half (51 participants) will receive rosuvastatin (the cholesterol lowering medication) and the other half (51 participants) will receive a placebo capsule. Participants will be recruited into the trial from two sites; here at the Alfred Hospital in Melbourne Australia and also from the University Hospital of Geneva in Switzerland. It is anticipated that 72 participants will be from Melbourne with the remaining 30 participants from Switzerland.

This project is a collaboration between the Infectious Diseases and Cardiology departments of the Alfred Hospital and the Infectious Diseases Department of the University Hospital of Geneva

#### 6 Do I have to take part in this research project?

Participation in any research project is voluntary. If you do not wish to take part, you do not have to. If you decide to take part and later change your mind, you are free to withdraw from the project at any stage.

Your decision whether to take part or not to take part, or to take part and then withdraw, will not affect your routine treatment, your relationship with those treating you or your relationship with the Alfred

#### 7 What are the alternatives to participation?

The use of rosuvastatin in people with normal cholesterol levels who are not at high risk for heart disease is experimental, and there is no standard clinical treatment which is similar or equal to this. Your alternative is to not join the study and continue to receive standard HIV care from your doctor.

#### 8 What are the possible benefits of taking part?

We cannot guarantee or promise that you will receive any benefits from your participation in this research. However the results from this research may help improve the management of people who are infected with HIV.

By participating in this study the health of your arteries and risk for heart problems will be assessed very thoroughly, in some instances this may allow us to detect serious treatable health issues before you have symptoms.

#### 9 What are the possible risks and disadvantages of taking part?

Medical treatments often cause side effects. You may have none, some or all of the effects listed below, and they may be mild, moderate or severe. If you have any of these side effects, or are worried about them, talk with your study doctor. Your study doctor will also be looking out for side effects.

There may be side effects that the researchers do not expect or do not know about and that may be serious. Tell your study doctor immediately about any new or unusual symptoms that you get.

Many side effects go away shortly after treatment ends. However, sometimes side effects can be serious, long lasting or permanent. If a severe side effect or reaction occurs, your study doctor may need to stop your treatment. Your study doctor will discuss the best way of managing any side effects with you.

Rosuvastatin is in general a safe medication that has been taken by many patients worldwide. Some side effects that can be caused by rosuvastatin include

- Muscle problems. Rosuvastatin can very occasionally (less than 1 per 1000 patients)
  cause serious muscle problems that can lead to kidney problems, including kidney
  failure and rarely, death.
- Liver problems. Rosuvastatin can occasionally cause liver problems that may rarely be serious or cause death. Your study nurse or doctor will do blood tests to check your liver before you start taking rosuvastatin, and while you take it.

Be sure to let your doctor or study nurse know immediately if you have possible signs of one of these problems, including:

- Muscle problems like weakness, tenderness, or pain that happen without a good reason, especially if you also have a fever or feel more tired than usual.
- Nausea and vomiting.

- o Passing brown or dark-colored urine.
- Feeling more tired than usual.
- o Noticing the skin and whites of your eyes become yellow.
- Having stomach pain.

Other problems that have been caused by rosuvastatin include headaches, rash, severe allergic reaction or swelling, constipation, gas, diarrhea, tendon rupture, dizziness, memory impairment, and depression. All these problems are uncommon to rare (occurring in less than 1 in 100 people who take rosuvastatin).

Having a blood sample taken may cause some discomfort, bruising, minor infection or bleeding. If this happens, it can be easily treated.

If, during the course of the study we uncover a medical condition that you did not know about the study doctor will explain the condition and arrange for you to have any further investigations or treatment that is necessary.

If you develop any condition (such as high cholesterol) which means that you should be taking rosuvastatin you will not be able to continue in the study and will be advised to stop taking the study medication and to take treatment as recommended by your usual doctor.

Study information that is not critical to your health care will not be given to you or others. This means that no one (not you, your family, your GP, your insurance company or your employer) will have access to this information during the study. At the end of the study you and your GP will be provided with a summary of the results of the study and your personal results including cholesterol levels and estimated risk of developing heart disease in the future.

#### Risks related to conception, pregnancy and breast feeding

Rosuvastatin is unsafe for unborn babies. Because of this, it is important that research project participants are not pregnant or breast-feeding and do not become pregnant during the course of the research project. You must not participate in the research if you are pregnant or trying to become pregnant, or breast-feeding. If you are female and child-bearing is a possibility, you will be required to undergo a pregnancy test prior to commencing the research project. If you are male, you should not father a child or donate sperm for at least one month after the last dose of study medication.

Both male and female participants are strongly advised to use effective contraception during the course of the research and for one month after completion of the research project. You should discuss methods of effective contraception with your study doctor.

If you do become pregnant whilst participating in the research project, you should advise your study doctor immediately. Your study doctor will withdraw you from the research project and advise on further medical attention should this be necessary. You must not continue in the research if you become pregnant.

You should advise your study doctor if you father a child while participating in the research project. Your study doctor will advise on medical attention for your partner should this be necessary.

If you become upset or distressed as a result of your participation in the research, the study doctor will be able to arrange for counselling or other appropriate support. Any counselling or

support will be provided by qualified staff who are not members of the research project team. This counselling will be provided free of charge.

#### 10 What will happen to my test samples?

By signing the consent form you are consenting to the collection of your blood for the research project.

The samples that you provide will not be used for any purpose other than what has been described in this document. Samples that are part of routine care will be tested at the Alfred Hospital and are destroyed as per hospital policy.

If you consent a small sample of blood will be stored for possible use in other research into the causes and prevention of heart disease in HIV and the actions of "statins". This may include (but is not limited to) testing for newly discovered markers of inflammation or performing special cholesterol studies. These samples would only be used for future research that has been approved by The Alfred Hospital Ethics Committee.

Your stored blood samples and the information collected about you during the study will be assigned a unique identifying code (that is not your name or birth date). This code will mean that results will be able to be re-identified and linked to individual study participants if needed. A small portion of your sample may be sent to Geneva for specialised testing. This sample will not have your name or date of birth on it and will be labelled only with the study code described above. There will be no need to take any extra blood samples and only samples from participants who have consented to having blood stored for future research will be included. If this does occur any blood remaining after testing is complete in Geneva will be destroyed.

The images taken with the ultrasound machine of the arteries in your neck will be stored on a CD and sent to Montreal, Canada where a specialist will review them, This CD will be labelled with the study code assigned to you and, as with your blood samples, will not contain your name or date of birth. At the completion of the trial the CD will be destroyed and your images will only be retained on file at the Alfred Hospital.

#### 11 What if new information arises during this research project?

Sometimes during the course of a research project, new information becomes available about the treatment that is being studied. If this happens, your study doctor will tell you about it and discuss with you whether you want to continue in the research project. If you decide to withdraw, your study doctor will make arrangements for your regular health care to continue. If you decide to continue in the research project you will be asked to sign an updated consent form.

Also, on receiving new information, your study doctor might consider it to be in your best interests to withdraw you from the research project. If this happens, he/ she will explain the reasons and arrange for your regular health care to continue.

#### 12 Can I have other treatments during this research project?

It is important to tell your study doctor and the study staff about any treatments or medications you may be taking, including over-the-counter medications, vitamins or herbal remedies, acupuncture or other alternative treatments. You should also tell your study doctor about any changes to these during your participation in the research project.

#### 13 What if I withdraw from this research project?

If you decide to withdraw from the project, please notify a member of the research team before you withdraw. This notice will allow that person or the research supervisor to discuss any health risks or special requirements linked to withdrawing.

If you do withdraw your consent during the research project, the study doctor and relevant study staff will not collect additional personal information from you, although personal information already collected will be retained to ensure that the results of the research project can be measured properly and to comply with law. You should be aware that data collected up to the time you withdraw will form part of the research project results, unless you specifically request otherwise.

#### 14 Could this research project be stopped unexpectedly?

It is not anticipated that this project will be stopped unexpectedly. However, this research project may be stopped early if unacceptable side effects were detected.

#### 15 What happens when the research project ends?

After you have completed all the study visits you will stop taking the study medication.

You and your GP will be sent a letter summarising your personal results including cholesterol levels and estimated risk of developing heart disease in the future. Once the whole study is finished you will receive a short report summarising the main findings of the study.

#### Part 2 How is the research project being conducted?

#### 16 What will happen to information about me?

By signing the consent form you consent to the study doctor and relevant research staff collecting and using personal information about you for the research project. Any information obtained in connection with this research project that can identify you will remain confidential. Information and samples will not be labelled with your name but will instead be assigned a code that will enable them to be re-identified and linked to individual study participants. This will be essential to perform the required study analyses and to monitor for potential side effects. Your information will only be used for the purpose of this research project and it will only be disclosed with your permission, except as required by law.

Information about you may be obtained from your health records held at The Alfred Hospital for the purpose of this research. By signing the consent form you agree to the study team accessing health records if they are relevant to your participation in this research project.

All research records will be kept in locked files located within locked rooms to which only study staff have access. Computer files will be stored on secure password protected computers

Only study staff, members of The Alfred Hospital Ethics Committee and regulatory authorities will have access to study data and participant information. The data and samples will not be used for commercial purposes. Written information will be retained indefinitely according to Alfred Health policy unless you ask for data to be destroyed.

It is anticipated that the results of this research project will be published and presented in a variety of forums. In any publication or presentation, information will be provided in such a way that you cannot be identified, except with your permission.

Information about your participation in this research project may be recorded in your health records.

In accordance with relevant Australian and Victorian privacy and other relevant laws, you have the right to request access to your information collected and stored by the research team. You also have the right to request that any information with which you disagree be corrected. Please contact the study team member named at the end of this document if you would like to access your information.

#### 17 Complaints and compensation

If you suffer any injuries or complications as a result of this research project, you should contact the study team as soon as possible and you will be assisted with arranging appropriate medical treatment. If you are eligible for Medicare, you can receive any medical treatment required to treat the injury or complication, free of charge, as a public patient in any Australian public hospital.

#### 18 Who is organising and funding the research?

This research project is being conducted by Professor Jennifer Hoy

You will not benefit financially from your involvement in this research project even if, for example, your samples (or knowledge acquired from analysis of your samples) prove to be of commercial value to The Alfred Hospital.

No member of the research team will receive a personal financial benefit from your involvement in this research project (other than their ordinary wages).

#### 19 Who has reviewed the research project?

All research in Australia involving humans is reviewed by an independent group of people called a Human Research Ethics Committee (HREC). The ethical aspects of this research project have been approved by the HREC of The Alfred Hospital Ethics Committee and the ethics committee the University Hospital of Geneva

This project will be carried out according to the *National Statement on Ethical Conduct in Human Research (2007)*. This statement has been developed to protect the interests of people who agree to participate in human research studies.

#### 20 Further information and who to contact

The person you may need to contact will depend on the nature of your guery.

If you want any further information concerning this project or if you have any medical problems which may be related to your involvement in the project (for example, any side effects), you can contact the principal study doctor on 90762000 or any of the following people:

### Clinical contact person

| Name | Dr Janine Trevillyan |
|-----------|-----------------------------------------------------|
| Position | Study co-ordinator and principal researcher |
| Telephone | 03 90762000 via Alfred Switchboard (24 hours a day) |
| Email | j.trevillyan@alfred.org.au |

| Name | Sally Price |
|-----------|----------------------------|
| Position | Study co-ordinator |
| Telephone | 03 9076 6908 |
| Email | clinresearch@alfred.org.au |

If you have any complaints about any aspect of the project, the way it is being conducted or any questions about being a research participant in general, then you may contact:

### **Complaints contact person**

| Name | Ms Rowan Frew |
|-----------|----------------------|
| Position | Ethics Manager |
| Telephone | 90763848 |
| Email | r.frew@alfred.org.au |

#### **Consent Form**

Title Does Rosuvastatin delay progression of atherosclerosis

in people with HIV infection? A multicentre randomized.

double blind placebo-controlled trial

**Coordinating Principal** 

Investigator/ Principal Investigator

Prof Jennifer Hov Associate Investigator(s)

Professor Suzanne Crowe

Dr Janine Trevillyan

Dr Julian Elliott

A. Professor Anthony Jaworowski

Dr James Shaw

Professor Anthony Dart

Location The Alfred Hospital

#### **Declaration by Participant**

I have read the Participant Information Sheet or someone has read it to me in a language that I understand.

I understand the purposes, procedures and risks of the research described in the project.

I give permission for my doctors, other health professionals, hospitals or laboratories outside this hospital to release information to The Alfred Hospital concerning my disease and treatment for the purposes of this project. I understand that such information will remain confidential.

I have had an opportunity to ask questions and I am satisfied with the answers I have received.

I freely agree to participate in this research project as described and understand that I am free to withdraw at any time during the study without affecting my future health care.

| I understand that I will be given a signed copy of this document to keep. | |
|---|---|
| Name of Participant (please | |
| Signature | Date |
| Name of Witness* to | |
| Participant's Signature (please print) | |
| Signature | Date |

#### Declaration by Study Doctor/Senior Researchert

I have given a verbal explanation of the research project, its procedures and risks and I believe that the participant has understood that explanation.

<sup>\*</sup> Witness is not to be the investigator, a member of the study team or their delegate. In the event that an interpreter is used, the interpreter may not act as a witness to the consent process. Witness must be 18 years or older.

| Name of Study Doctor/ Senior Researcher† (please print) | |
|---|---|
| Signature | Date |
| | mber of the research team must provide the explanation of, and information ne research project. |
| Note: All parti | es signing the consent section must date their own signature. |
| Consent for storage and use of blood samples | |
| Please indicat | e your choice by checking (ticking) ONE of the options below: |
| | I consent to the use of my blood samples for tests related to this research |
| | project <u>and</u> for a sample to be stored for future research as described in the relevant section of the Participant information sheet |
| <u>OR</u> | relevant section of the Farticipant information sheet |
| | I consent to the use of blood samples taken from me for use in this project as |
| | described in the relevant section of the Participant Information Sheet but <u>do</u> <u>not</u> authorize their future use in any other research. |
| Name of I | Participant (please |
| Signature | Date |
| | Witness* to t's Signature (please |
| Signature | Date |
| event that an | ot to be the investigator, a member of the study team or their delegate. In the interpreter is used, the interpreter may <u>not</u> act as a witness to the consent ness must be 18 years or older. |
| | Study Doctor/<br>esearcher <sub>t</sub> (please |
| Signature | Date |

<sup>†</sup> A senior member of the research team must provide the explanation of and information concerning the research project.

Note: All parties signing the consent section must date their own signature
## Form for Withdrawal of Participation - Adult providing own consent

**Title** Does Rosuvastatin delay progression of atherosclerosis

in people with HIV infection? A multicentre randomized,

double blind placebo-controlled trial

**Coordinating Principal** 

Investigator/ Principal Investigator

Dr Janine Trevillyan Prof Jennifer Hoy

Associate Investigator(s) Professor Suzanne Crowe

Dr Julian Elliott

A. Professor Anthony Jaworowski

Dr James Shaw

**Professor Anthony Dart** 

**Location** The Alfred Hospital

## **Declaration by Participant**

Signature

I wish to withdraw from participation in the above research project and understand that such withdrawal will not affect my routine treatment, my relationship with those treating me or my relationship with The Alfred Hospital

| Name of Participant (please | |
|---|---|
| Signature | Date |
| · | on to withdraw is communicated verbally, the Study rovide a description of the circumstances below. |
| Declaration by Study Doctor/Senior R | esearcher <sub>t</sub> |
| I have given a verbal explanation of the idea and I believe that the participant has unc | implications of withdrawal from the research project derstood that explanation. |
| Name of Study Doctor/ Senior Researcher <sub>†</sub> (please print) | |

\_\_\_\_\_ Date \_\_\_\_

<sup>&</sup>lt;sup>+</sup> A senior member of the research team must provide the explanation of and information concerning withdrawal from the research project. Note: All parties signing the consent section must date their own signature.

## 22.6 Severity Grading of Adverse Events

# Modified DIVISION OF AIDS TABLE FOR GRADING THE SEVERITY OF ADULT ADVERSE EVENTS

VERSION 1.0, DECEMBER, 2004; CLARIFICATION AUGUST 2009

The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events ("DAIDS AE Grading Table") is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term.

### **Instructions and Clarifications**

In the classification of adverse events, the term "severe" is not the same as "serious." Severity is an indication of the intensity of a specific event (as in mild, moderate, or severe chest pain). The term "serious" relates to a participant/event outcome or action criteria, usually associated with events that pose a threat to a participant's life or functioning.

For any AE where the outcome is death, the severity of the AE is classified as Grade 5.

Determining Severity Grade for Parameters "Between Grades"

If the severity of a clinical AE could fall under either one of two grades (e.g., the severity of an AE could be either Grade 2 or Grade 3), select the higher of the two grades for the AE. If a laboratory value that is graded as a multiple of the ULN or LLN falls between two grades, select the higher of the two grades for the AE. For example, Grade 1 is 2.5 x ULN and Grade 2 is 2.6 x ULN for a parameter. If the lab value is

2.53 x ULN (which is between the two grades), the severity of this AE would be Grade 2, the higher of the two grades.

Values Below Grade 1: Any laboratory value that is between either the LLN or ULN and Grade 1 should not be graded.

### **Definitions of terms used in the Table:**

Basic Self-care Functions Activities such as bathing, dressing, toileting,

transfer/movement, continence, and feeding

LLN Lower limit of normal

Medical Intervention Use of pharmacologic or biologic agent(s) for treatment

of an AE.

NA Not Applicable

Operative Intervention Surgical OR other invasive mechanical procedures

ULN Upper limit of normal

| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|
| ESTIMATING SEVERITY GRADE | | | | |
| Clinical adverse event<br>NOT identified<br>elsewhere in this<br>DAIDS AE Grading<br>Table | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Symptoms causing inability to perform basic self-care functions OR Medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death |
| SYSTEMIC | | | | |
| Acute systemic allergic reaction | Localized urticaria<br>(wheals) with no<br>medical intervention<br>indicated | Localized urticaria with medical intervention indicated OR Mild angioedema with no medical intervention indicated | Generalized urticaria<br>OR Angioedema with<br>medical intervention<br>indicated OR<br>Symptomatic mild<br>bronchospasm | Acute anaphylaxis OR<br>Life-threatening<br>bronchospasm OR<br>laryngeal edema |
| Chills | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | NA |
| Fatigue<br>Malaise | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Incapacitating fatigue/<br>malaise symptoms<br>causing inability to<br>perform basic self-care<br>functions |
| Fever (nonaxillary) | 37.7 – 38.6°C | 38.7 – 39.3°C | 39.4 – 40.5°C | > 40.5°C |
| Pain (indicate body<br>site) DO NOT use for pain<br>due to injection (See<br>Injection Site<br>Reactions: Injection<br>site pain) See also Headache,<br>Arthralgia, and<br>Myalgia | Pain causing no or minimal interference with usual social & functional activities | Pain causing greater<br>than minimal<br>interference with usual<br>social & functional<br>activities | Pain causing inability to perform usual social & functional activities | Disabling pain causing inability to perform basic self-care functions OR Hospitalization (other than emergency room visit) indicated |
| Unintentional weight loss | NA | 5 – 9% loss in body<br>weight from baseline | 10 – 19% loss in body<br>weight from baseline | 20% loss in body weight<br>from baseline OR<br>Aggressive intervention<br>indicated [e.g., tube<br>feeding or total<br>parenteral nutrition<br>(TPN)] |

| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|
| INFECTION | | | | |
| Infection (any other<br>than HIV infection) | Localized, no<br>systemic antimicrobial<br>treatment indicated<br>AND Symptoms<br>causing no or minimal<br>interference with<br>usual social &<br>functional activities | Systemic antimicrobial treatment indicated OR Symptoms causing greater than minimal interference with usual social & functional activities | Systemic antimicrobial treatment indicated AND Symptoms causing inability to perform usual social & functional activities OR Operative intervention (other than simple incision and drainage) indicated | Life-threatening<br>consequences (e.g.,<br>septic shock) |
| INJECTION SITE RE | ACTIONS | | | |
| Injection site pain<br>(pain without touching)<br>Or<br>Tenderness (pain<br>when area is touched) | Pain/tenderness<br>causing no or minimal<br>limitation of use of<br>limb | Pain/tenderness<br>limiting use of limb OR<br>Pain/tenderness<br>causing greater than<br>minimal interference<br>with usual social &<br>functional activities | Pain/tenderness<br>causing inability to<br>perform usual social &<br>functional activities | Pain/tenderness causing inability to perform basic self-care function OR Hospitalization (other than emergency room visit) indicated for management of pain/tenderness |
| Injection site reaction (localized) | Erythema OR<br>Induration<br>of 5x5 cm – 9x9 cm<br>(or 25 cm <sup>2</sup> – 81cm <sup>2</sup> ) | Erythema OR<br>Induration OR Edema<br>> 9 cm any diameter<br>(or > 81 cm <sup>2</sup> ) | Ulceration OR<br>Secondary infection OR<br>Phlebitis OR Sterile<br>abscess OR Drainage | Necrosis (involving dermis and deeper tissue) |
| Pruritis associated with injection See also Skin: Pruritis (itching - no skin lesions) | Itching localized to injection site AND Relieved spontaneously or with < 48 hours treatment | Itching beyond the injection site but not generalized OR Itching localized to injection site requiring 48 hours treatment | Generalized itching causing inability to perform usual social & functional activities | N/A |
| SKIN - DERMATOL | OGICAL | | | |
| Alopecia | Thinning detectable by study participant (or by caregiver for young children and disabled adults) | Alopecia | Thinning detectable by study participant (or by caregiver for young children and disabled adults) | Alopecia |
| Cutaneous reaction (Rash) | Localized macular rash | Diffuse macular,<br>maculopapular, or<br>morbilliform rash OR<br>Target lesions | maculopapular, or<br>morbilliform rash with<br>vesicles or limited<br>number of bullae OR<br>Superficial ulcerations<br>of mucous membrane<br>limited to one site | Extensive or generalized bullous lesions OR Stevens-Johnson syndrome OR Ulceration of mucous membrane involving two or more distinct mucosal sites OR Toxic epidermal necrolysis (TEN) |
| Pruritis (itching – no<br>skin lesions)<br>(See also Injection Site<br>Reactions: Pruritis<br>associated with<br>injection) | minimal interference with usual social & functional | Itching causing greater<br>than minimal interference<br>with usual social &<br>functional activities | Itching causing inability<br>to perform usual social<br>& functional activities | NA |

| Vasovagal episode<br>(associated with a<br>procedure of any kind) | Present without loss of consciousness | Present with transient loss of consciousness | NA | NA |
|---|---|---|---|---|
| Ventricular dysfunction (congestive heart failure) | NA | Asymptomatic diagnostic finding AND intervention indicated | New onset with symptoms OR Worsening symptomatic congestive heart failure | Life-threatening congestive heart failure |
| GASTROINTESTINAL | | | | |
| Anorexia | Loss of appetite without decreased oral intake | Loss of appetite<br>associated with<br>decreased oral intake<br>without significant<br>weight loss | Loss of appetite associated with significant weight loss | Life-threatening consequences OR Aggressive intervention indicated [e.g., tube feeding or total parenteral nutrition (TPN)] |
| Ascites | Asymptomatic | Symptomatic AND<br>Intervention indicated<br>(e.g., diuretics or<br>therapeutic<br>paracentesis) | Symptomatic despite intervention | Life-<br>threatening<br>consequence<br>s |
| Cholecystitis | NA | Symptomatic AND<br>Medical intervention<br>indicated | Radiologic,<br>endoscopic,or operative<br>intervention indicated | Life-threatening consequences (e.g., sepsis or perforation) |
| Constipation | NA | Persistent constipation requiring regular use of dietary modifications, laxatives, or enemas | Obstipation with manual evacuation indicated | Life-threatening consequences (e.g., obstruction) |
| Diarrhea | Transient or intermittent episodes of unformed stools OR Increase of ≤ 3 stools over baseline per 24-hour period | Persistent episodes of<br>unformed to watery<br>stools OR Increase of<br>4 – 6 stools over<br>baseline per 24-hour<br>period | Bloody diarrhea OR<br>Increase of ≥7 stools<br>per 24-hour period OR<br>IV fluid replacement<br>indicated | Life-threatening<br>consequences<br>(e.g., hypotensive<br>shock) |
| Dysphagia-<br>Odynophagia | Symptomatic but able to eat usual diet | Symptoms causing altered dietary intake without medical intervention indicated | Symptoms causing severely altered dietary intake with medical intervention indicated | Life-threatening<br>reduction in oral<br>intake |

| Mucositis/stomatitis (clinical exam) Indicate site (e.g., larynx, oral) See Genitourinary for Vulvovaginitis | Erythema of the mucosa | Patchy pseudomembranes or ulcerations | Confluent pseudomembranes or ulcerations OR Mucosal bleeding with minor trauma | Tissue necrosis OR Diffuse spontaneous mucosal bleeding OR Life- threatening consequences |
|---|---|---|---|---|
| Nausea | Transient (< 24 hours) or intermittent nausea with no or minimal interference with oral intake | Persistent nausea<br>resulting in decreased<br>oral intake for 24 – 48<br>hours | Persistent nausea<br>resulting in minimal oral<br>intake for > 48 hours<br>OR Aggressive<br>rehydration indicated<br>(e.g., IV fluids) | Life-threatening<br>consequences<br>(e.g., hypotensive<br>shock) |

| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|
| Pancreatitis | NA | Symptomatic AND<br>Hospitalization not<br>indicated (other than<br>emergency room visit) | Symptomatic AND<br>Hospitalization indicated<br>(other than emergency<br>room visit) | Life-threatening<br>consequences (e.g.,<br>circulatory failure,<br>hemorrhage, sepsis) |
| Proctitis (functional-<br>symptomatic)<br>Also see<br>Mucositis/stomatitis<br>for clinical exam | Rectal discomfort<br>AND No intervention<br>indicated | Symptoms causing greater than minimal interference with usual social & functional activities OR Medical intervention indicated | Symptoms causing inability to perform usual social & functional activities OR Operative intervention indicated | Life-threatening consequences (e.g., perforation) |
| Vomiting | Transient or intermittent vomiting with no or minimal interference with oral intake | Frequent episodes of vomiting with no or mild dehydration | Persistent vomiting resulting in orthostatic hypotension OR Aggressive rehydration indicated (e.g., IV fluids) | Life-threatening<br>consequences (e.g.,<br>hypotensive shock) |
| NEUROLOGIC | | | | |
| Alteration in personality-behavior or in mood (e.g., agitation, anxiety, depression, mania, psychosis) | Alteration causing no or minimal interference with usual social & functional activities | Alteration causing greater than minimal interference with usual social & functional activities | Alteration causing inability to perform usual social & functional activities | Behavior potentially harmful to self or others (e.g., suicidal and homicidal ideation or attempt, acute psychosis) OR Causing inability to perform basic self-care functions |
| Altered Mental Status For Dementia, see Cognitive and behavioral/attentional disturbance (including dementia and attention deficit disorder) | Changes causing no or minimal interference with usual social & functional activities | Mild lethargy or<br>somnolence causing<br>greater than minimal<br>interference with usual<br>social & functional<br>activities | Confusion, memory impairment, lethargy, or somnolence causing inability to perform usual social & functional activities | Delirium OR obtundation, OR coma |

| Ataxia Cognitive and | Asymptomatic ataxia detectable on exam OR Minimal ataxia causing no or minimal interference with usual social & functional activities Disability causing no or | Symptomatic ataxia causing greater than minimal interference with usual social & functional activities Disability causing greater | Symptomatic ataxia causing inability to perform usual social & functional activities Disability causing inability | Disabling ataxia causing inability to perform basic self-care functions Disability causing inability to |
|---|---|---|---|---|
| behavioral/attentional disturbance (including | minimal interference with usual social & functional activities OR Specialized | than minimal interference<br>with usual social &<br>functional activities OR<br>Specialized resources on<br>part-time basis indicated | to perform usual social & functional activities OR Specialized resources on a full-time basis indicated | perform basic self-care functions OR Institutionalization indicated |
| CNS ischemia<br>(acute) | NA | NA | Transient ischemic attack | Cerebral vascular accident<br>(CVA, stroke) with<br>neurological deficit |
| Headache | Symptoms causing no or<br>minimal<br>interference with usual<br>social &<br>functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Symptoms causing inability to perform basic self-care functions OR Hospitalization indicated (other than emergency room visit) OR Headache with significant impairment of alertness or other neurologic function |
| Insomnia | NA | Difficulty sleeping causing<br>greater than minimal<br>interference with usual<br>social & functional<br>activities | Difficulty sleeping causing inability to perform usual social & functional activities | Disabling insomnia causing inability to perform basic self-care functions |
| Neuromuscular<br>weakness<br>(including myopathy & | Asymptomatic with decreased strength on exam OR Minimal muscle weakness causing no or minimal interference with usual social & functional activities | greater than minimal interference with usual social & functional activities Muscle weakness causing greater than minimal | inability to perform usual social & functional activities | inability to perform basic |
| Neuromuscular<br>weakness<br>(including myopathy & | Asymptomatic with decreased strength on exam OR Minimal muscle weakness causing no or minimal interference with usual social & | greater than minimal interference with usual social & functional activities Muscle weakness causing greater than minimal interference with usual social & functional | inability to perform usual social & functional activities Muscle weakness causing inability to perform usual social & functional | inability to perform basic self-care functions Disabling muscle weakness causing inability to perform basic self-care functions OR Respiratory muscle weakness impairing |

| NA | Increased frequency of pre-existing seizures (non-repetitive) without change in seizure character OR Infrequent break- through seizures while on stable medication in a previously controlled seizure disorder | Change in seizure character from baseline either in duration or quality (e.g., severity or focality) | Seizures of any kind<br>which are prolonged,<br>repetitive (e.g., status<br>epilepticus), or difficult<br>to control (e.g.,<br>refractory epilepsy) |
|---|---|---|---|
| Vertigo causing no or minimal interference with usual social & functional activities | Vertigo causing greater<br>than minimal<br>interference with usual<br>social & functional<br>activities | Vertigo causing inability to perform usual social & functional activities | Disabling vertigo causing inability to perform basic self-care functions |
| GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| FEV1 or peak flow<br>reduced to<br>70 – 80% | FEV1 or peak flow<br>50 <b>–</b> 69% | FEV1 or peak flow<br>25 <b>–</b> 49% | Cyanosis OR FEV1 or peak flow < 25% OR Intubation |
| Dyspnea on exertion with no or minimal interference with usual social & functional activities | Dyspnea on exertion causing greater than minimal interference with usual social & functional activities | Dyspnea at rest causing inability to perform usual social & functional activities | Respiratory failure with ventilatory support indicated |
| AL | | | |
| Joint pain causing no or minimal interference with usual social & functional activities | Joint pain causing greater than minimal interference with usual social & functional activities | Joint pain causing inability to perform usual social & functional activities | Disabling joint pain causing inability to perform basic self-care functions |
| Stiffness or joint swelling causing no or minimal interference with usual social & functional activities | Stiffness or joint swelling causing greater than minimal interference with usual social & functional activities | Stiffness or joint<br>swelling causing<br>inability to perform usual<br>social & functional<br>activities | Disabling joint stiffness or<br>swelling causing inability<br>to perform basic self-care<br>functions |
| BMD t-score<br>-2.5 to -1.0 | BMD t-score < -2.5 | Pathological fracture (including loss of vertebral height) | Pathologic fracture causing life-threatening consequences |
| Muscle pain causing no or minimal interference with usual social & functional activities | Muscle pain causing greater than minimal interference with usual social & functional activities | Muscle pain causing inability to perform usual social & functional activities | Disabling muscle pain causing inability to perform basic self-care functions |
| NA | Asymptomatic with radiographic findings AND No operative intervention indicated | Symptomatic bone pain with radiographic findings OR Operative intervention indicated | Disabling bone pain with radiographic findings causing inability to perform basic self-care functions |
| | Vertigo causing no or minimal interference with usual social & functional activities GRADE 1 MILD FEV1 or peak flow reduced to 70 – 80% Dyspnea on exertion with no or minimal interference with usual social & functional activities AL Joint pain causing no or minimal interference with usual social & functional activities Stiffness or joint swelling causing no or minimal interference with usual social & functional activities BMD t-score -2.5 to -1.0 Muscle pain causing no or minimal interference with usual social & functional activities | pre-existing seizures (non-repetitive) without change in seizure character OR Infrequent break- through seizures while on stable medication in a previously controlled seizure disorder Vertigo causing no or minimal interference with usual social & functional activities GRADE 1 | pre-existing seizures (non-repetitive) without change in seizure character OR Infrequent break-through seizures while on stable medication in a previously controlled seizure disorder |

| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|
| GENITOURINARY | | | | |
| Cervicitis<br>(symptoms)<br>(For use in studies<br>evaluating topical<br>study agents) | Symptoms causing or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Symptoms causing inability to perform basic self-care functions |
| Cervicitis (clinical exam) (For use in studies evaluating topical study agents) For other cervicitis see Infection: Infection (any other than HIV infection) | Minimal cervical abnormalities on examination (erythema, mucopurulent discharge, or friability) OR Epithelial disruption | Moderate cervical abnormalities on examination (erythema, mucopurulent discharge, or friability) OR Epithelial disruption of 25 – 49% total surface | Severe cervical<br>abnormalities on<br>examination (erythema,<br>mucopurulent<br>discharge, or friability)<br>OR Epithelial disruption<br>50 – 75% total surface | Epithelial disruption > 75% total surface |
| Inter-menstrual bleeding (IMB) | Spotting observed participant OR Minimal blood observed during clinical or colposcopic examination | Inter-menstrual<br>bleeding not greater in<br>duration or amount<br>than usual menstrual<br>cycle | Inter-menstrual bleeding<br>greater in duration or<br>amount than usual<br>menstrual cycle | Hemorrhage with life-<br>threatening hypotension<br>OR Operative<br>intervention indicated |
| Urinary tract<br>obstruction (e.g.,<br>stone) | N | Signs or symptoms of<br>urinary tract<br>obstruction without<br>hydronephrosis or<br>renal dysfunction | Signs or symptoms of urinary tract obstruction with hydronephrosis or renal dysfunction | Obstruction causing life-<br>threatening<br>consequences |
| OCULAR/VISUAL | | | | |
| Uveitis | Asymptomatic but detectable on exam | Symptomatic<br>anterior uveitis OR<br>Medical<br>intervention | Posterior or pan-uveitis<br>OR Operative<br>intervention indicated | Disabling visual loss in affected eye(s) |
| Visual changes (from baseline) | Visual changes causing no or minimal interference with usual social & functional activities | Visual changes causing greater than minimal interference with usual social & functional activities | Visual changes causing inability to perform usual social & functional activities | Disabling visual loss in affected eye(s) |
| ENDOCRINE/METAE | ENDOCRINE/METABOLIC | | | |
| Abnormal fat accumulation (e.g., back of neck, breasts, abdomen) | Detectable by study<br>participant (or by<br>caregiver for young<br>children and disabled<br>adults) | Detectable on physica exam by health care provider | Disfiguring OR Obvious changes on casual visual inspection | NA |

| Diabetes mellitus | NA | New onset without need to initiate medication OR Modification of current medications to regain glucose | New onset with initiation of medication indicated OR Diabetes uncontrolled despite treatment modification | Life-threatening<br>consequences (e.g.,<br>ketoacidosis,<br>hyperosmolar non-<br>ketotic coma) |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Gynecomastia | Detectable by study participant or caregiver (for young children and disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious on casual visual inspection | NA |
| Hyperthyroidism | Asymptomatic | Symptomatic causing greater than minimal interference with usual social & functional activities OR Thyroid suppression therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life-threatening consequences (e.g., thyroid storm) |
| Hypothyroidism | Asymptomatic | Symptomatic causing greater than minimal interference with usual social & functional activities OR Thyroid replacement therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life-threatening consequences (e.g., myxedema coma) |
| Lipoatrophy<br>(e.g., fat loss from<br>the face,<br>extremities,<br>buttocks) | Detectable by study participant (or by caregiver for young children and disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious on casual visual inspection | NA |

| LABORATORY | | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| HEMATOLOGY | Standard Internationa | I Units are listed in ita | alics | |
| Absolute neutrophil count (ANC) | 1.000 x 10 <sup>9</sup> –<br>1.300 x 10 <sup>9</sup> /L | 0.750 x 10 <sup>9</sup> –<br>0.999 x 10 <sup>9</sup> /L | 0.500 x 10 <sup>9</sup> –<br>0.749 x 10 <sup>9</sup> /L | < 0.500 x 10 <sup>9</sup> /L |
| Fibrinogen, decreased | 1.00 – 2.00 g/L<br>OR<br>0.75 – 0.99 x LLN | 0.75 – 0.99 g/L<br>OR<br>0.50 – 0.74 x LLN | 0.50 – 0.74 g/L<br>OR<br>0.25 – 0.49 x LLN | < 0.50 g/L<br>OR<br>< 0.25 x LLN<br>OR<br>Associated with gross<br>bleeding |

| | LABORATORY | | | |
|---|---|---|---|---|
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Hemoglobin (Hgb) | <u>,L,</u> | | | |
| HIV POSITIVE ONLY | 8.5 – 10.0 g/dL | 7.5 – 8.4 g/dL | 6.50 – 7.4 g/dL | < 6.5 g/dL |
| HIV NEGATIVE<br>ONLY | 10.0 – 10.9 g/dL<br>OR<br>Any decrease<br>2.5 – 3.4 g/dL | 9.0 – 9.9 g/dL<br>OR<br>Any decrease<br>3.5 – 4.4 g/dL | 7.0 – 8.9 g/dL<br>OR<br>Any decrease<br>ε4.5 g/dL | < 7.0 g/dL |
| Comment: The decrease | is a decrease from baselin | ne | | |
| International Normalized<br>Ratio of prothrombin time<br>(INR) | 1.1 – 1.5 x ULN | 1.6 – 2.0 x ULN | 2.1 – 3.0 x ULN | > 3.0 x ULN |
| Methemoglobin | 5.0 – 10.0% | 10.1 – 15.0% | 15.1 – 20.0% | > 20.0% |
| Prothrombin Time (PT) | 1.1 – 1.25 x ULN | 1.26 – 1.50 x ULN | 1.51 – 3.00 x ULN | > 3.00 x ULN |
| Partial Thromboplastin<br>Time (PTT) | 1.1 – 1.66 x ULN | 1.67 – 2.33 x ULN | 2.34 – 3.00 x ULN | > 3.00 x ULN |
| Platelets, decreased | 100.000 x 10 <sup>9</sup> –<br>124.999 x 10 <sup>9</sup> /L | 50.000 x 10 <sup>9</sup> –<br>99.999 x 10 <sup>9</sup> /L | 25.000 x 10 <sup>9</sup> –<br>49.999 x 10 <sup>9</sup> /L | < 25.000 x 10 <sup>9</sup> /L |
| WBC, decreased | 2.000 x 10 <sup>9</sup> –<br>2.500 x 10 <sup>9</sup> /L | 1.500 x 10 <sup>9</sup> –<br>1.999 x 10 <sup>9</sup> /L | 1.000 x 10 <sup>9</sup> –<br>1.499 x 10 <sup>9</sup> /L | < 1.000 x 10 <sup>9</sup> /L |
| CHEMISTRIES | | | <u> </u> | |
| Acidosis | NA | pH < normal, but ε7.3 | pH < 7.3 without life-<br>threatening<br>consequences | pH < 7.3 with life-<br>threatening<br>consequences |
| Albumin, serum, low | 30 g/L - < LLN | 20 – 29 g/L | < 20 g/L | NA |
| Alkaline Phosphatase | 1.25 – 2.5 x ULN <sup>†</sup> | 2.6 – 5.0 x ULN <sup>†</sup> | 5.1 – 10.0 x ULN <sup>†</sup> | > 10.0 x ULN <sup>†</sup> |
| Alkalosis | NA | pH > normal, but δ7.5 | pH > 7.5 without life-<br>threatening<br>consequences | pH > 7.5 with life-<br>threatening<br>consequences |
| ALT (SGPT) | 1.25 – 2.5 x ULN | 2.6 – 5.0 x ULN | 5.1 – 10.0 x ULN | > 10.0 x ULN |
| AST (SGOT) | 1.25 – 2.5 x ULN | 2.6 – 5.0 x ULN | 5.1 – 10.0 x ULN | > 10.0 x ULN |
| Bicarbonate, serum, low | 16.0 mmol/L – < LLN | 11.0 – 15.9 mmol/L | 8.0 – 10.9 mmol/L | < 8.0 mmol/L |
| Bilirubin (Total) | 1.1 – 1.5 x ULN | 1.6 – 2.5 x ULN | 2.6 – 5.0 x ULN | > 5.0 x ULN |
| Calcium, serum, high | 2.65 – 2.88 mmol/L | 2.89 – 3.13 mmol/L | 3.14 – 3.38 mmol/L | > 3.38 mmol/L |
| Calcium, serum, low | 1.95 – 2.10 mmol/L | 1.75 – 1.94 mmol/L | 1.53 – 1.74 mmol/L | < 1.53 mmol/L |

| Cardiac troponin I (cTnI) | NA | NA | | Levels consistent with myocardial infarction or unstable angina as defined by the manufacturer |
|---|---|---|---|---|
| Creatine Kinase | 3.0 – 5.9 x ULN† | 6.0 – 9.9 x ULN† | 10.0 – 19.9 x ULN† | ≥□20.0 x ULN† |
| Creatinine | 1.1 – 1.3 x ULN† | 1.4 – 1.8 x ULN† | 1.9 – 3.4 x ULN† | ≥□3.5 x ULN† |

| Lipase | 1.1 – 1.5 x ULN | 1.6 – 3.0 x ULN | 3.1 – 5.0 x ULN | > 5.0 x ULN |
|---|---|---|---|---|
| Lactate | ULN - < 2.0 x ULN without acidosis | ε2.0 x ULN without acidosis | Increased lactate with pH < 7.3 without life- | Increased lactate with pH < 7.3 with life- |
| Magnesium, serum, low | 0.60 – 0.70 mmol/L | 0.45 – 0.59 mmol/L | 0.30 – 0.44 mmol/L | < 0.30 mmol/L |
| Pancreatic amylase | 1.1 – 1.5 x ULN | 1.6 – 2.0 x ULN | 2.1 – 5.0 x ULN | > 5.0 x ULN |
| Phosphate, serum, low | 0.81 mmol/L - < LLN | 0.65 – 0.80 mmol/L | 0.32 – 0.64 mmol/L | < 0.32 mmol/L |
| Potassium, serum, high | 5.6 – 6.0 mmol/L | 6.1 – 6.5 mmol/L | 6.6 – 7.0 mmol/L | > 7.0 mmol/L |
| Potassium, serum, low | 3.0 – 3.4 mmol/L | 2.5 – 2.9 mmol/L | 2.0 – 2.4 mmol/L | < 2.0 mmol/L |
| Sodium, serum, high | 146 – 150 mmol/L | 151 – 154 mmol/L | 155 – 159 mmol/L | ε160 mmol/L |
| Sodium, serum, low | 130 – 135 mmol/L | 125 – 129 mmol/L | 121 – 124 mmol/L | δ120 mmol/L |
| URINALYSIS Standard International Units are listed in italics | | | | |
| Hematuria (microscopic) | 6 – 10 RBC/HPF | > 10 RBC/HPF | Gross, with or without clots OR with RBC casts | Transfusion indicated |
| Proteinuria, random collection | 1+ | 2-3+ | 4+ | NA |
| Proteinuria, 24 hour colle | ection | • | | • |
| Adult | 0.200 – 0.999 g/d | 1.000 – 1.999 g/d | 2.000 - 3.500 g/d | > 3.500 g/d |
| | • | · | | • |

| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|
| Glucose, serum, high | | | | |
| Nonfasting | 6.44 – 8.88 mmol/L | 8.89 – 13.88 mmol/L | 13.89 – 27.75 mmol/L | > 27.75 mmol/L |
| Fasting | 6.11 – 6.94 mmol/L | 6.95 – 13.88 mmol/L | 13.89 – 27.75 mmol/L | > 27.75 mmol/L |
| Glucose, serum, low | 3.05 – 3.55 mmol/L | 2.22 – 3.06 mmol/L | 1.67 – 2.23 mmol/L | < 1.67 mmol/L |